CLINICAL TRIAL: NCT05184452
Title: A Phase 1 Dose-escalation Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of PGDM1400LS Alone and in Combination With VRC07-523LS and PGT121.414.LS in Healthy, HIV-uninfected Adult Participants
Brief Title: A Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of PGDM1400LS Alone and in Combination With VRC07-523LS and PGT121.414.LS in Healthy, HIV-uninfected Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 140/HPTN 101; DAIDS DOCUMENT ID (Other: 38723)
Record Dates: First submitted 2021-10-26; First posted 2022-01-11 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- PGDM1400LS 5 mg/kg IV (Experimental): Participants will receive PGDM1400LS 5 mg/kg by intravenous (IV) infusion at Month 0
  Interventions: Drug: PGDM1400LS (5mg/kg, IV)
- PGDM1400LS 20 mg/kg IV (Experimental): Participants will receive PGDM1400LS 20 mg/kg by IV infusion at Month 0
  Interventions: Drug: PGDM1400LS (20mg/kg, IV)
- PGDM1400LS 20 mg/kg SC (Experimental): Participants will receive PGDM1400LS 20 mg/kg by subcutaneous (SC) infusion at Month 0
  Interventions: Drug: PGDM1400LS (20mg/kg, SC)
- PGDM1400LS 40 mg/kg IV (Experimental): Participants will receive PGDM1400LS 40 mg/kg by IV infusion at Month 0
  Interventions: Drug: PGDM1400LS (40mg/kg, IV)
- PGDM1400LS 40 mg/kg SC (Experimental): Participants will receive PGDM1400LS 40 mg/kg by SC infusion at Month 0
  Interventions: Drug: PGDM1400LS (40mg/kg, SC)
- PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg IV (Experimental): Participants will receive PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg by IV infusion sequentially in this order at Month 0 and Month 4
  Interventions: Drug: PGDM1400LS (20mg/kg, IV); Drug: VRC07-523LS (20mg/kg, IV); Drug: PGT121.414.LS (20mg/kg, IV)
- PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg SC (Experimental): Participants will receive PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg by SC infusion sequentially in this order at Month 0 and Month 4
  Interventions: Drug: PGDM1400LS (20mg/kg, SC); Drug: VRC07-523LS (20mg/kg, SC); Drug: PGT121.414.LS (20mg/kg, SC)
- PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram IV (Experimental): Participants will receive PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram by IV infusion sequentially in this order at Month 0 and Month 4
  Interventions: Drug: PGDM1400LS (1.4g, IV); Drug: VRC07-523LS (1.4g, IV); Drug: PGT121.414.LS (1.4g, IV)
- PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram SC (Experimental): Participants will receive PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram by SC infusion sequentially in this order at Month 0 and Month 4
  Interventions: Drug: PGDM1400LS (1.4g, SC); Drug: VRC07-523LS (1.4g, SC); Drug: PGT121.414.LS (1.4g, SC)
- PGDM1400LS 40mg/kg + VRC07-523LS 40mg/kg + PGT121.414.LS 40 mg/kg IV (Experimental): Participants will receive PGDM1400LS 40mg/kg + VRC07-523LS 40mg/kg + PGT121.414.LS 40 mg/kg by IV infusion sequentially in this order at Month 0 and Month 4
  Interventions: Drug: PGDM1400LS (40mg/kg, IV); Drug: VRC07-523LS (40mg/kg, IV); Drug: PGT121.414.LS (40mg/kg, IV)

INTERVENTIONS:
Drug: PGDM1400LS (5mg/kg, IV) — 5 mg/kg to be administered via IV infusion
  Arms: PGDM1400LS 5 mg/kg IV
Drug: PGDM1400LS (20mg/kg, IV) — 20 mg/kg to be administered via IV infusion
  Arms: PGDM1400LS 20 mg/kg IV; PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg IV
Drug: PGDM1400LS (20mg/kg, SC) — 20 mg/kg to be administered via SC infusion
  Arms: PGDM1400LS 20 mg/kg SC; PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg SC
Drug: PGDM1400LS (40mg/kg, IV) — 40 mg/kg to be administered via IV infusion
  Arms: PGDM1400LS 40 mg/kg IV; PGDM1400LS 40mg/kg + VRC07-523LS 40mg/kg + PGT121.414.LS 40 mg/kg IV
Drug: PGDM1400LS (40mg/kg, SC) — 40 mg/kg to be administered via SC infusion
  Arms: PGDM1400LS 40 mg/kg SC
Drug: PGDM1400LS (1.4g, IV) — 1.4gram to be administered via IV infusion
  Arms: PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram IV
Drug: PGDM1400LS (1.4g, SC) — 1.4gram to be administered via SC infusion
  Arms: PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram SC
Drug: VRC07-523LS (20mg/kg, IV) — VRC07-523LS 20mg/kg administered via IV infusion
  Arms: PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg IV
Drug: VRC07-523LS (20mg/kg, SC) — VRC07-523LS 20mg/kg administered via SC infusion
  Arms: PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg SC
Drug: VRC07-523LS (1.4g, IV) — VRC07-523LS 1.4g administered via IV infusion
  Arms: PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram IV
Drug: VRC07-523LS (1.4g, SC) — VRC07-523LS 1.4g administered via SC infusion
  Arms: PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram SC
Drug: VRC07-523LS (40mg/kg, IV) — VRC07-523LS 40mg/kg administered via IV infusion
  Arms: PGDM1400LS 40mg/kg + VRC07-523LS 40mg/kg + PGT121.414.LS 40 mg/kg IV
Drug: PGT121.414.LS (20mg/kg, IV) — PGT121.414.LS 20mg/kg administered via IV infusion
  Arms: PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg IV
Drug: PGT121.414.LS (20mg/kg, SC) — PGT121.414.LS 20mg/kg administered via SC infusion
  Arms: PGDM1400LS 20mg/kg + VRC07-523LS 20mg/kg + PGT121.414.LS 20 mg/kg SC
Drug: PGT121.414.LS (1.4g, IV) — PGT121.414.LS 1.4g administered via IV infusion
  Arms: PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram IV
Drug: PGT121.414.LS (1.4g, SC) — PGT121.414.LS 1.4g administered via SC infusion
  Arms: PGDM1400LS 1.4gram + VRC07-523LS 1.4gram + PGT121.414.LS 1.4gram SC
Drug: PGT121.414.LS (40mg/kg, IV) — PGT121.414.LS 40mg/kg administered via IV infusion
  Arms: PGDM1400LS 40mg/kg + VRC07-523LS 40mg/kg + PGT121.414.LS 40 mg/kg IV

SUMMARY:
Part A:

The purpose of this part of the study is to understand how the body's immune system responds to a new lab-made antibody against HIV. The study is looking to see if the way the antibody is given affects the immune response. The study will also look at whether the antibody is safe to give to people and does not make them too uncomfortable.

Part B:

The purpose of this part of the study is to understand how the body's immune system responds to lab-made antibodies against HIV when they are given in combination at different doses. The study also wants to see if the way the antibodies are given affects the immune response.

DETAILED DESCRIPTION:
The HIV Vaccine Trials Network (HVTN) and the HIV Prevention Trials Network (HPTN) are conducting this study to test a combination of different antibodies against HIV. HIV is the virus that causes AIDS. Antibodies are made by the body as one way to respond to or fight infection. Researchers can also make antibodies in laboratories and give them to people by infusions into a vein or under the skin.

There are 2 parts of this study, Part A and Part B. About 15 people will take part in Part A of this study to test one study antibody. After early safety results from Part A are obtained, a decision will be made as to whether or not to do Part B of the study. Part B of the study would test a combination of 3 antibodies. If it is decided to move forward with Part B, 80 more people will join.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 through 50 years
2. Access to a participating CRS and willingness to be followed for the planned duration of the study
3. Ability and willingness to provide informed consent
4. Assessment of understanding: volunteer demonstrates understanding of this study and completes a questionnaire prior to first study product administration with verbal demonstration of understanding of all questionnaire items answered incorrectly
5. Agrees not to enroll in another study of an investigational research agent until completion of the last required protocol clinic visit.
6. Good general health as shown by medical history, physical exam, and screening laboratory tests
7. Willingness to receive HIV test results
8. Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
9. Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit (see Appendix J and Appendix K).
10. Hemoglobin

    * ≥ 11.0 g/dL for volunteers who were assigned female sex at birth
    * ≥ 13.0 g/dL for volunteers who were assigned male sex at birth and transgender males who have been on hormone therapy for more than 6 consecutive months
    * ≥ 12.0 g/dL for transgender females who have been on hormone therapy for more than 6 consecutive months
    * For transgender volunteers who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on the sex assigned at birth
11. White blood cell count = 2,500 to 12,000 cells/mm3
12. WBC differential either within institutional normal range or with site clinician approval
13. Platelets = 125,000 to 550,000 cells/mm3
14. Chemistry panel: alanine aminotransferase (ALT) < 1.25 times the institutional upper limit of normal (ie, < 1.25 times the reference range upper limit) and creatinine < 1.1 times the institutional upper limit of normal (ie, <1.1 times the reference range upper limit)
15. Negative HIV-1 and -2 blood test: US volunteers must have a negative FDA-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA). Non-US sites may use locally available assays that have been approved by HVTN and HPTN Laboratory Operations
16. Negative Hepatitis B surface antigen (HBsAg)
17. Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
18. Negative or trace urine protein
19. Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test(s) performed within 48 hours prior to initial study product administration. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
20. A volunteer who was assigned female sex at birth must:

    * Agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol visit. Effective contraception is defined as using one of the following methods: Condoms (internal and external) with or without a spermicide, Diaphragm or cervical cap with spermicide, Intrauterine device (IUD), Hormonal contraception, Tubal ligation, or Any other contraceptive method approved by the HVTN 140/HPTN 101 PSRT, Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy); or,
    * Not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy or bilateral oophorectomy; or,
    * Be sexually abstinent.
21. Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

1. Weight < 35kg or > 115 kg
2. Blood products received within 120 days before first study product administration, unless eligibility for earlier enrollment is determined by the HVTN 140/HPTN 101 PSRT
3. Investigational research agents received within 30 days before first study product administration
4. Intent to participate in another study of an investigational research agent or any other study that requires non-Network HIV antibody testing during the planned duration of the HVTN 140/HPTN 101 study
5. Pregnant or breastfeeding
6. HIV vaccine(s) received in a prior HIV vaccine trial. Volunteers who have received control/placebo in an HIV vaccine trial are not excluded.
7. SARS-CoV-2 vaccine(s) received within 7 days prior to HVTN 140/HPTN 101 enrollment or planned within 7 days after enrollment.
8. Receipt of humanized or human mAbs, whether licensed or investigational.
9. Previous receipt of mAbs VRC01, VRC01LS, VRC07-523LS, PGDM1400, PGT121, PGT121.414.LS.
10. Immunosuppressive medications received within 30 days before first study product administration (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatological condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses < 20 mg/day and length of therapy < 14 days)
11. Serious adverse reactions to PGDM1400LS, VRC07-523LS, or PGT121.414.LS formulation components (see Section 8.2) including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
12. Immunoglobulin received within 60 days before first study product administration (for mAb see criterion 8 above)
13. Autoimmune disease (Not excluded from participation: Volunteer with mild, stable and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgment of the CRS investigator, is likely not subject to exacerbation and likely not to complicate Solicited and Unsolicited AE assessments.)
14. Immunodeficiency
15. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    * Symptoms consistent with COVID-19 or known SARS-CoV-2 infection,
    * A process that would affect the immune response,
    * A process that would require medication that affects the immune response,
    * Any contraindication to repeated infusions, or blood draws, including inability to establish venous or subcutaneous access,
    * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
    * A condition or process (eg, chronic urticaria or recent injection or infusion with evidence of residual inflammation) for which signs or symptoms could be confused with reactions to the study product, or
    * Any condition specifically listed among the exclusion criteria.
16. Any medical, psychiatric, or skin condition (eg, tattoos), or occupational responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of safety or Solicited AEs, or a participant's ability to give informed consent.
17. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
18. Current anti-tuberculosis (TB) therapy
19. Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).

    Exclude a volunteer who:
    * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
    * Uses moderate/high-dose, inhaled corticosteroids, or
    * In the past year has had either of the following: Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids; Emergency care, urgent care, hospitalization, or intubation for asthma.
20. Diabetes mellitus type 1 or type 2 (Not excluded: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
21. Hypertension:

    * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined in this protocol as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
    * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
22. Bleeding disorder diagnosed by a clinician (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
23. Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
24. Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
25. Asplenia: any condition resulting in the absence of a functional spleen
26. History of generalized urticaria, angioedema, or anaphylaxis (Not exclusionary: angioedema or anaphylaxis to a known trigger with at least 5 years since last reaction to demonstrate satisfactory avoidance of trigger).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, Study Chair — Emory University; Marc Siegel, Study Chair — George Washington University; Sharana Mahomed, Study Chair — Centre for the AIDS Programme of Research in South Africa
Locations (13):
- United States (5):
  - Bridge HIV CRS, San Francisco, California
  - George Washington University, Washington D.C., District of Columbia
  - The Hope Clinic of the Emory Vaccine Center, Atlanta, Georgia
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Vanderbilt Vaccine (VV), Nashville, Tennessee
- Kenya Medical Research Institute (KEMRI), Kericho, Kenya
- South Africa (4):
  - CAPRISA eThekweni Clinical Research Site, Berea, Durban
  - Ward 21 Clinical Research Site, Hillbrow, Johannesburg
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Soweto HVTN CRS, Soweto
- Zimbabwe (3):
  - Seke South Clinical Research Site, Chitungwiza, Harare
  - Milton Park CRS, Milton Park, Harare
  - Spilhaus CRS, Milton Park, Harare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seaton KE, Paez CA, Yu C, Karuna ST, Gamble T, Miner MD, Heptinstall J, Zhang L, Gao F, Yacovone M, Spiegel H, Dumond JB, Anderson M, Piwowar-Manning E, Dye B, Tindale I, Proulx-Burns L, Trahey M, Takuva S, Takalani A, Bailey VC, Kalams SA, Scott H, Mkhize NN, Weiner JA, Ackerman ME, McElrath MJ, Pensiero M, Barouch DH, Montefiori D, Tomaras GD, Corey L, Cohen MS, Huang Y, Mahomed S, Siegel M, Kelley CF; HVTN 140/HPTN 101 study team. Safety, pharmacokinetics, and neutralisation activity of PGDM1400LS, a V2 specific HIV-1 broadly neutralising antibody, infused intravenously or subcutaneously in people without HIV-1 in the USA (HVTN 140/HPTN 101 part A): a first-in-human, phase 1 randomised trial. Lancet HIV. 2025 Jun;12(6):e405-e415. doi: 10.1016/S2352-3018(25)00012-8. PMID 40441807

RESULTS

PARTICIPANT FLOW:
Groups:
- T1: PGDM1400LS (IV) 5 mg/kg mo 0: PGDM1400LS 5 mg/kg to be administered IV at Month 0.
- T2: PGDM1400LS (IV) 20 mg/kg mo 0: PGDM1400LS 20 mg/kg to be administered IV at Month 0.
- T3: PGDM1400LS (SC) 20 mg/kg mo 0: PGDM1400LS 20 mg/kg to be administered SC at Month 0.
- T4: PGDM1400LS (IV) 40 mg/kg mo 0: PGDM1400LS 40 mg/kg to be administered IV at Month 0.
- T5: PGDM1400LS (SC) 40 mg/kg mo 0: PGDM1400LS 40 mg/kg to be administered SC at Month 0.
- T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2: PGDM1400LS 20 mg/kg AND VRC07-523LS 20 mg/kg AND PGT121.414LS 20 mg/kg to be administered IV sequentially in this order at Month 0 and Month 4.
- T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2: PGDM1400LS 20 mg/kg AND VRC07-523LS 20 mg/kg AND PGT121.414LS 20 mg/kg to be administered SC sequentially in this order at Month 0 and Month 4.
- T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1: PGDM1400LS 1.4 g AND VRC07-523LS 1.4 g AND PGT121.414LS 1.4 g to be administered IV sequentially in this order at Month 0 and Month 4.
- T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1: PGDM1400LS 1.4 g AND VRC07-523LS 1.4 g AND PGT121.414LS 1.4 g to be administered SC sequentially in this order at Month 0 and Month 4.
- T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV): PGDM1400LS 40 mg/kg AND VRC07-523LS 40 mg/kg AND PGT121.414LS 40 mg/kg to be administered IV sequentially in this order at Month 0 and Month 4.
Period: Overall Study
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Started | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
Completed | 3 | 3 | 3 | 3 | 3 | 13 | 16 | 16 | 16 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16 | 95
Age, Continuous [Median (Full Range); unit: years] | 36 [25 to 38] | 27 [24 to 27] | 27 [25 to 34] | 26 [24 to 32] | 33 [29 to 47] | 25.5 [18 to 46] | 27.5 [18 to 46] | 25.5 [18 to 45] | 26 [18 to 48] | 31 [19 to 45] | 27 [18 to 48]
Age, Customized [Count of Participants; unit: Participants]
  18 - 20 years | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 3 | 2 | 12
  21 - 30 years | 1 | 3 | 2 | 2 | 1 | 9 | 9 | 7 | 8 | 4 | 46
  31 - 40 years | 2 | 0 | 1 | 1 | 1 | 2 | 3 | 2 | 2 | 7 | 21
  41 - 50 years | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 3 | 3 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 2 | 9 | 9 | 9 | 6 | 5 | 48
  Male | 1 | 1 | 1 | 1 | 1 | 7 | 7 | 7 | 10 | 11 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 6
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 2 | 14 | 15 | 15 | 16 | 15 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 12 | 13 | 11 | 13 | 10 | 60
  White | 1 | 3 | 2 | 3 | 2 | 4 | 2 | 3 | 2 | 4 | 26
  More than one race | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 6 | 4 | 6 | 38
  Kenya | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 3 | 0 | 9
  South Africa | 0 | 0 | 0 | 0 | 0 | 8 | 7 | 8 | 6 | 4 | 33
  Zimbabwe | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 3 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured through Month Measured through 3 days after each vaccine dose at T1-T5: Day 0 and T6-T10: Days 0, 112
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
Participants
  None | 3 | 2 | 2 | 3 | 2 | 15 | 9 | 13 | 3 | 14
  Mild | 0 | 1 | 1 | 0 | 1 | 1 | 6 | 3 | 12 | 2
  Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through Month Measured through 3 days after each vaccine dose at T1-T5: Day 0 and T6-T10: Days 0, 112
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
Participants
  Erythema/Redness: None | 3 | 3 | 2 | 3 | 1 | 16 | 12 | 16 | 10 | 16
  Erythema/Redness: Mild | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Erythema/Redness: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 0
  Erythema/Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: None | 3 | 3 | 2 | 3 | 1 | 16 | 13 | 16 | 10 | 16
  Induration/Swelling: Mild | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
  Induration/Swelling: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Induration/Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 3 | 3 | 2 | 3 | 1 | 16 | 12 | 16 | 9 | 16
  Erythema and/or Induration: Mild | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
  Erythema and/or Induration: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through Month Measured through 3 days after each vaccine dose at T1-T5: Day 0 and T6-T10: Days 0, 112
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
Participants
  Malaise and/or fatigue: None | 3 | 1 | 3 | 2 | 3 | 9 | 10 | 9 | 11 | 13
  Malaise and/or fatigue: Mild | 0 | 2 | 0 | 1 | 0 | 5 | 5 | 4 | 5 | 1
  Malaise and/or fatigue: Moderate | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 1
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 3 | 3 | 3 | 3 | 3 | 13 | 12 | 12 | 14 | 13
  Myalgia: Mild | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 2
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 3 | 1 | 2 | 2 | 2 | 7 | 10 | 10 | 12 | 10
  Headache: Mild | 0 | 1 | 1 | 1 | 1 | 6 | 6 | 3 | 4 | 4
  Headache: Moderate | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 2
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 2 | 3 | 3 | 3 | 3 | 11 | 15 | 14 | 12 | 14
  Nausea: Mild | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 3 | 2
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 3 | 3 | 3 | 3 | 3 | 12 | 16 | 13 | 14 | 14
  Chills: Mild | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 2
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 3 | 3 | 3 | 3 | 3 | 13 | 16 | 15 | 13 | 14
  Arthralgia: Mild | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 2
  Arthralgia: Moderate | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Facial flushing: None | 3 | 3 | 3 | 3 | 3 | 15 | 15 | 16 | 15 | 16
  Facial flushing: Mild | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Facial flushing: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Facial flushing: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Facial flushing: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional dyspnea: None | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 15 | 16 | 16
  Non-exertional dyspnea: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Non-exertional dyspnea: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional dyspnea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional dyspnea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional tachycardia: None | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
  Non-exertional tachycardia: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unexplained diaphoresis: None | 3 | 3 | 3 | 3 | 3 | 12 | 16 | 15 | 16 | 16
  Unexplained diaphoresis: Mild | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Unexplained diaphoresis: Moderate | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Unexplained diaphoresis: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unexplained diaphoresis: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: None | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 15 | 16 | 16
  Generalized Pruritus: Mild | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Generalized Pruritus: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: None | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
  Urticaria: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 2 | 1 | 2 | 2 | 2 | 7 | 7 | 6 | 7 | 10
  Max. Systemic Symptoms: Mild | 1 | 1 | 1 | 1 | 1 | 5 | 8 | 5 | 8 | 3
  Max. Systemic Symptoms: Moderate | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 5 | 1 | 2
  Max. Systemic Symptoms: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 15
  Temperature: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP)
Description: For each local laboratory measure, summary statistics: median and interquartile range were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during Screening, Days 0, 56, 112*, 168, and 280* Days with * are only available for T6-T10
Population: 'Overall Number of Participants Analyzed' represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
U/L
  ALP (U/L) -Day 0/Enrollment | 62 [30 to 71] | 56 [53 to 76] | 73 [43 to 86] | 73 [71 to 96] | 78 [68 to 91] | 76.5 [61.5 to 107] | 73.5 [61.5 to 104] | 75 [61 to 85] | 85 [70 to 118.5] | 72 [62 to 87.5]
  ALP (U/L) -Day 56: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  ALP (U/L) -Day 56 | 40.5 [32 to 49] | 65 [51 to 81] | 68 [45 to 79] | 75 [74 to 86] | 59 [59 to 79] | 77 [55 to 101] | 68.5 [65.5 to 95.5] | 74.5 [65.5 to 91.5] | 81.5 [67 to 107] | 83 [70 to 89]
  ALP (U/L) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 14
  ALP (U/L) -Day 112 |  |  |  |  |  | 77 [59 to 97] | 72 [65 to 107] | 70.5 [56 to 96] | 84 [67.5 to 109] | 76 [65 to 102]
  ALP (U/L) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  ALP (U/L) -Day 168 | 48 [33 to 55] | 63 [47 to 88] | 72 [40 to 90] | 84 [71 to 88] | 81 [72 to 89] | 83.5 [62 to 104] | 74 [72 to 101.5] | 73 [71 to 93] | 84 [64.5 to 102] | 78 [67 to 91]
  ALP (U/L) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  ALP (U/L) -Day 280 |  |  |  |  |  | 73 [61 to 111] | 78 [64 to 84] | 72 [60 to 83] | 86.5 [68.5 to 97.5] | 76 [64 to 97]
  AST (U/L) -Day 0/Enrollment | 19 [17 to 26] | 16 [14 to 18] | 21 [14 to 22] | 20 [16 to 20] | 21 [13 to 25] | 21 [18 to 26] | 20.5 [17 to 24.5] | 18 [16 to 21.5] | 24 [16 to 29] | 20.5 [17 to 24]
  AST (U/L) -Day 56: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  AST (U/L) -Day 56 | 17.5 [16 to 19] | 15 [15 to 19] | 21 [16 to 22] | 20 [19 to 22] | 21 [14 to 22] | 21 [19 to 29] | 19 [16.5 to 23] | 18.5 [17 to 25] | 24 [21 to 29] | 21 [17 to 30]
  AST (U/L) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 14
  AST (U/L) -Day 112 |  |  |  |  |  | 20.5 [19 to 30] | 20 [16 to 22] | 18.5 [16.5 to 27] | 24 [19 to 27] | 24.5 [17 to 42]
  AST (U/L) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  AST (U/L) -Day 168 | 16 [15 to 48] | 19 [14 to 23] | 19 [14 to 19] | 20 [16 to 20] | 23 [13 to 24] | 22.5 [20 to 26] | 22.5 [20 to 27.5] | 23.5 [17 to 25] | 25 [17.5 to 29] | 20 [16 to 28]
  AST (U/L) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  AST (U/L) -Day 280 |  |  |  |  |  | 23 [17 to 28] | 21 [18 to 25.5] | 18.5 [16 to 22] | 22.5 [19 to 27.5] | 21 [18 to 24]
  ALT (U/L) -Screening: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 15 | 16
  ALT (U/L) -Screening | 15 [10 to 20] | 14 [7 to 28] | 15 [10 to 19] | 17 [12 to 25] | 18 [9 to 25] | 16.5 [12.5 to 23.5] | 13.5 [9.5 to 16.5] | 16.5 [11.5 to 27] | 14 [11 to 19] | 15 [11.5 to 25]
  ALT (U/L) -Day 0/Enrollment | 14 [14 to 17] | 16 [6 to 28] | 12 [12 to 27] | 17 [10 to 18] | 16 [12 to 29] | 19.5 [13 to 22.5] | 13 [10 to 17] | 16 [10.5 to 21] | 14 [11 to 19] | 18.5 [12.5 to 26.5]
  ALT (U/L) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  ALT (U/L) -Day 56 | 16 [14 to 18] | 13 [8 to 23] | 12 [10 to 26] | 18 [14 to 20] | 15 [14 to 26] | 19 [15 to 22] | 13 [10 to 16.5] | 16 [12.5 to 24] | 17.5 [14 to 23.5] | 18 [12 to 25]
  ALT (U/L) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 14
  ALT (U/L) -Day 112 |  |  |  |  |  | 21 [12 to 34] | 14 [9 to 20] | 16 [14 to 24] | 18.5 [13.5 to 23] | 16 [14 to 32]
  ALT (U/L) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  ALT (U/L) -Day 168 | 15 [10 to 34] | 16 [7 to 33] | 10 [8 to 23] | 14 [12 to 16] | 14 [13 to 54] | 18.5 [15 to 32] | 16 [12 to 23] | 17 [14 to 30] | 17 [11 to 25] | 16.5 [12 to 36]
  ALT (U/L) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  ALT (U/L) -Day 280 |  |  |  |  |  | 22 [11 to 29] | 13.5 [11.5 to 24.5] | 14.5 [12 to 20.5] | 15.5 [11.5 to 23] | 17.5 [13 to 30]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during Screening, Days 0, 56, 112*, 168, and 280* Days with * are only available for T6-T10
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
mg/dL
  Creatinine (mg/dL) -Screening | 0.77 [0.68 to 0.77] | 0.78 [0.74 to 0.87] | 0.83 [0.56 to 0.85] | 0.94 [0.89 to 1.03] | 0.81 [0.69 to 0.95] | 0.79 [0.64 to 0.85] | 0.72 [0.59 to 0.8] | 0.79 [0.66 to 0.9] | 0.79 [0.71 to 0.89] | 0.81 [0.69 to 0.92]
  Creatinine (mg/dL) -Day 0/Enrollment | 0.75 [0.74 to 0.8] | 0.79 [0.65 to 0.87] | 0.81 [0.64 to 0.99] | 0.85 [0.83 to 0.89] | 0.9 [0.72 to 0.91] | 0.8 [0.64 to 0.91] | 0.74 [0.65 to 0.81] | 0.7 [0.66 to 0.88] | 0.81 [0.77 to 0.89] | 0.82 [0.71 to 0.96]
  Creatinine (mg/dL) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Creatinine (mg/dL) -Day 56 | 0.81 [0.81 to 0.82] | 0.78 [0.67 to 1.02] | 0.8 [0.78 to 0.98] | 0.89 [0.76 to 0.91] | 0.82 [0.75 to 0.96] | 0.74 [0.65 to 0.83] | 0.7 [0.59 to 0.86] | 0.76 [0.72 to 0.83] | 0.77 [0.69 to 0.93] | 0.79 [0.67 to 0.94]
  Creatinine (mg/dL) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 14
  Creatinine (mg/dL) -Day 112 |  |  |  |  |  | 0.73 [0.59 to 0.84] | 0.74 [0.61 to 0.84] | 0.76 [0.68 to 0.83] | 0.79 [0.7 to 0.87] | 0.8 [0.7 to 0.88]
  Creatinine (mg/dL) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Creatinine (mg/dL) -Day 168 | 0.8 [0.77 to 0.83] | 0.83 [0.67 to 1.01] | 0.81 [0.74 to 1.09] | 0.89 [0.86 to 1.03] | 0.92 [0.73 to 0.96] | 0.73 [0.68 to 0.87] | 0.74 [0.66 to 0.85] | 0.74 [0.69 to 0.84] | 0.8 [0.72 to 0.94] | 0.81 [0.68 to 0.91]
  Creatinine (mg/dL) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Creatinine (mg/dL) -Day 280 |  |  |  |  |  | 0.74 [0.68 to 0.85] | 0.76 [0.6 to 0.89] | 0.81 [0.7 to 0.94] | 0.84 [0.7 to 0.89] | 0.78 [0.71 to 0.91]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin
Description: as for outcome 5
Time Frame: Measured during Screening, Days 0, 56, 112*, 168, and 280* Days with * are only available for T6-T10
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
g/dL
  Hemoglobin (g/dL) -Screening | 13.6 [12.7 to 14.8] | 14.3 [12.3 to 15.5] | 15.1 [12.3 to 16.7] | 13.3 [13.3 to 16.2] | 14.3 [12.6 to 14.5] | 14.5 [13.8 to 16.05] | 14.05 [13.35 to 14.6] | 14.1 [13.45 to 15.55] | 14.8 [13.35 to 15.55] | 15.8 [14.1 to 17.1]
  Hemoglobin (g/dL) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  Hemoglobin (g/dL) -Day 0/Enrollment | 12.3 [11.7 to 12.9] | 12.3 [11.8 to 15.1] | 13.7 [13.1 to 17.3] | 12.7 [11.5 to 16] | 13.6 [12.7 to 15] | 14.75 [14.2 to 16.75] | 13.5 [13.2 to 15.2] | 13.9 [12.6 to 15.7] | 14.35 [13.6 to 15.3] | 14.9 [13.5 to 16.75]
  Hemoglobin (g/dL) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Hemoglobin (g/dL) -Day 56 | 12.9 [11.6 to 14.5] | 13.6 [11.7 to 15.2] | 13.3 [12.9 to 17.3] | 13.5 [12.5 to 15.8] | 13.5 [11.8 to 14.5] | 14.5 [13.9 to 15.3] | 13.85 [13.3 to 14.95] | 13.85 [12.9 to 15.35] | 14.9 [13.15 to 15.4] | 14.9 [13.9 to 17.2]
  Hemoglobin (g/dL) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  Hemoglobin (g/dL) -Day 112 |  |  |  |  |  | 14.3 [13.3 to 16.2] | 13.6 [13.4 to 15.1] | 14 [12.75 to 15.25] | 14.6 [12.8 to 15.5] | 15 [13.4 to 18]
  Hemoglobin (g/dL) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Hemoglobin (g/dL) -Day 168 | 12.5 [11.6 to 16.7] | 14.3 [11.5 to 14.7] | 13 [12.9 to 17.5] | 13.9 [12.1 to 16.3] | 13.8 [12.3 to 14.4] | 14.75 [13.5 to 16] | 13.95 [13.55 to 15.2] | 13.4 [13 to 14.7] | 14.35 [13.05 to 15.15] | 15.45 [13.9 to 17.4]
  Hemoglobin (g/dL) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Hemoglobin (g/dL) -Day 280 |  |  |  |  |  | 13.8 [13.2 to 15.5] | 13.85 [13.4 to 15.25] | 13.8 [12.85 to 16] | 13.85 [13.1 to 14.75] | 15.05 [13.9 to 16.8]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count
Description: as for outcome 5
Time Frame: Measured during Screening, Days 0, 56, 112*, 168, and 280* Days with * are only available for T6-T10
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
1000 cells/cubic mm
  Neutrophils (1000 cells/cubic mm) -Screening | 4.3 [3.31 to 5.06] | 2.88 [2.19 to 3.7] | 5.36 [3.9 to 5.79] | 3.6 [3.1 to 4.58] | 4.28 [3.7 to 4.4] | 3.5 [2.58 to 4.5] | 3.48 [2.59 to 4.31] | 3.54 [2.91 to 3.79] | 2.95 [2.09 to 4.25] | 3 [2.15 to 3.5]
  Neutrophils (1000 cells/cubic mm) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  Neutrophils (1000 cells/cubic mm) -Day 0/Enrollment | 2.88 [1.74 to 4.02] | 2.81 [2.61 to 3.03] | 5.2 [4.22 to 5.53] | 2.8 [2.5 to 4.28] | 3.68 [2.91 to 4.18] | 3.35 [2.55 to 3.81] | 2.25 [1.78 to 3.48] | 3.01 [2.33 to 3.77] | 3.27 [1.54 to 4.28] | 2.77 [2.32 to 3.98]
  Neutrophils (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Neutrophils (1000 cells/cubic mm) -Day 56 | 2.76 [2.48 to 3.47] | 2.68 [2.5 to 2.92] | 4.87 [3.9 to 5.09] | 4.7 [3 to 5.02] | 4.81 [4.22 to 5.18] | 2.66 [2.1 to 4.54] | 2.87 [2.27 to 4.14] | 3.28 [2.36 to 4.07] | 2.72 [1.82 to 5.02] | 3.13 [2.19 to 3.7]
  Neutrophils (1000 cells/cubic mm) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  Neutrophils (1000 cells/cubic mm) -Day 112 |  |  |  |  |  | 2.54 [1.87 to 3.8] | 2.54 [1.69 to 3.85] | 2.84 [2.4 to 3.5] | 2.57 [1.63 to 3.62] | 2.73 [2.47 to 3.27]
  Neutrophils (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Neutrophils (1000 cells/cubic mm) -Day 168 | 3.44 [2.01 to 3.61] | 2.32 [1.47 to 3.49] | 4.66 [3.29 to 4.9] | 4.16 [3.5 to 4.5] | 5.53 [2.58 to 7.71] | 2.65 [1.92 to 3.76] | 2.8 [1.93 to 3.59] | 3.39 [2.98 to 4.11] | 2.92 [1.68 to 4.53] | 2.77 [2.05 to 3.11]
  Neutrophils (1000 cells/cubic mm) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Neutrophils (1000 cells/cubic mm) -Day 280 |  |  |  |  |  | 2.05 [1.71 to 2.91] | 2.72 [2.17 to 4.25] | 3.38 [2.74 to 4.48] | 3.29 [2.13 to 4.11] | 2.76 [2.54 to 3.13]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, White Blood Cells (WBC)
Description: as for outcome 5
Time Frame: Measured during Screening, Days 0, 56, 112*, 168, and 280* Days with * are only available for T6-T10
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
1000 cells/cubic mm
  WBC (1000 cells/cubic mm) -Screening | 7100 [6800 to 7200] | 5300 [4600 to 6600] | 7600 [6800 to 9300] | 6300 [5500 to 6600] | 6700 [6100 to 7700] | 6475 [5160 to 7050] | 6330 [5280 to 7290] | 6040 [5020 to 6650] | 5555 [4985 to 7280] | 5515 [4750 to 6400]
  WBC (1000 cells/cubic mm) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  WBC (1000 cells/cubic mm) -Day 0/Enrollment | 5900 [4900 to 6900] | 5300 [4700 to 5800] | 7900 [7600 to 10100] | 5900 [4400 to 7300] | 6400 [5400 to 7700] | 6045 [4805 to 6840] | 5110 [3800 to 6640] | 5320 [4640 to 6400] | 5255 [4020 to 7160] | 5470 [4795 to 6945]
  WBC (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  WBC (1000 cells/cubic mm) -Day 56 | 5700 [5300 to 6100] | 5200 [4300 to 5200] | 8500 [6900 to 9200] | 7000 [5400 to 7500] | 7200 [6900 to 7300] | 5000 [4110 to 7400] | 5110 [4480 to 6960] | 5285 [4735 to 7515] | 5120 [4525 to 7315] | 5240 [4300 to 6330]
  WBC (1000 cells/cubic mm) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  WBC (1000 cells/cubic mm) -Day 112 |  |  |  |  |  | 4880 [3950 to 6700] | 5570 [3955 to 6400] | 5210 [4450 to 6075] | 5210 [4130 to 5840] | 5320 [4440 to 5900]
  WBC (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  WBC (1000 cells/cubic mm) -Day 168 | 5700 [4800 to 5800] | 4900 [3800 to 6000] | 6700 [5900 to 9100] | 6100 [6100 to 8000] | 8600 [5400 to 11200] | 5335 [4030 to 6400] | 5425 [4055 to 6700] | 5690 [4800 to 6440] | 5575 [4115 to 7200] | 5085 [3880 to 6300]
  WBC (1000 cells/cubic mm) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  WBC (1000 cells/cubic mm) -Day 280 |  |  |  |  |  | 4240 [3880 to 5900] | 5385 [4295 to 6805] | 5550 [4895 to 6895] | 5845 [4180 to 7170] | 5025 [4500 to 5540]
  Platelets (1000 cells/cubic mm) -Screening | 252000 [192000 to 257000] | 304000 [243000 to 416000] | 288000 [281000 to 310000] | 324000 [227000 to 326000] | 298000 [274000 to 313000] | 282000 [250000 to 291500] | 299000 [255500 to 347000] | 280000 [257000 to 332500] | 275500 [217500 to 329000] | 249000 [229500 to 281500]
  Platelets (1000 cells/cubic mm) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  Platelets (1000 cells/cubic mm) -Day 0/Enrollment | 207000 [190000 to 224000] | 281000 [247000 to 405000] | 283000 [270000 to 323000] | 288000 [210000 to 338000] | 317000 [278000 to 349000] | 286000 [254500 to 306500] | 285000 [237000 to 322000] | 265000 [233000 to 283000] | 266000 [221000 to 334000] | 241500 [216000 to 283000]
  Platelets (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Platelets (1000 cells/cubic mm) -Day 56 | 237000 [171000 to 256000] | 295000 [243000 to 435000] | 289000 [288000 to 362000] | 293000 [211000 to 309000] | 294000 [264000 to 346000] | 277000 [248000 to 310000] | 293000 [242500 to 318000] | 287000 [261500 to 336500] | 268000 [248000 to 357000] | 263000 [230000 to 277000]
  Platelets (1000 cells/cubic mm) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  Platelets (1000 cells/cubic mm) -Day 112 |  |  |  |  |  | 283500 [243000 to 301000] | 285500 [254000 to 317000] | 278500 [222500 to 302000] | 253500 [231000 to 355500] | 261000 [225000 to 302000]
  Platelets (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Platelets (1000 cells/cubic mm) -Day 168 | 213000 [208000 to 241000] | 296000 [256000 to 387000] | 283000 [278000 to 336000] | 306000 [231000 to 385000] | 399000 [261000 to 420000] | 276500 [259000 to 293000] | 300500 [244000 to 364000] | 265500 [242000 to 298000] | 298000 [251500 to 329000] | 251000 [220000 to 329000]
  Platelets (1000 cells/cubic mm) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Platelets (1000 cells/cubic mm) -Day 280 |  |  |  |  |  | 267000 [207000 to 290000] | 300000 [253000 to 346000] | 293500 [259000 to 340500] | 296500 [243500 to 327000] | 248000 [224000 to 325000]

9. Primary Outcome: Number of Lab Grade >= 1 for Alanine Aminotransferase (ALT), Creatinine, Hemoglobin, Lymphocyte Count, Neutrophil Count, Platelets, White Blood Cells (WBC).
Description: The number (percentage) of participants with lab grade >= 1 for alanine aminotransferase (ALT),Â creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC) was summarized by arm
Time Frame: Measured during Screening, Days 0, 56, 112*, 168, and 280* Days with * are only available for T6-T10
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
Participants
  ALP (U/L) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
  ALP (U/L) -Day 56: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  ALP (U/L) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  ALP (U/L) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 14
  ALP (U/L) -Day 112 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALP (U/L) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  ALP (U/L) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  ALP (U/L) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  ALP (U/L) -Day 280 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST (U/L) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L) -Day 56: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  AST (U/L) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  AST (U/L) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 14
  AST (U/L) -Day 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  AST (U/L) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  AST (U/L) -Day 168 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  AST (U/L) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  AST (U/L) -Day 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  ALT (U/L) -Screening: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 15 | 16
  ALT (U/L) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALT (U/L) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  ALT (U/L) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  ALT (U/L) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 14
  ALT (U/L) -Day 112 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3
  ALT (U/L) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  ALT (U/L) -Day 168 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 2
  ALT (U/L) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  ALT (U/L) -Day 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hemoglobin (g/dL) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  Hemoglobin (g/dL) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Hemoglobin (g/dL) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  Hemoglobin (g/dL) -Day 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Hemoglobin (g/dL) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Hemoglobin (g/dL) -Day 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Creatinine (mg/dL) -Day 56 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 14
  Creatinine (mg/dL) -Day 112 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Creatinine (mg/dL) -Day 168 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Creatinine (mg/dL) -Day 280 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  WBC (1000 cells/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  WBC (1000 cells/cubic mm) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  WBC (1000 cells/cubic mm) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  WBC (1000 cells/cubic mm) -Day 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  WBC (1000 cells/cubic mm) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  WBC (1000 cells/cubic mm) -Day 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  Platelets (1000 cells/cubic mm) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Platelets (1000 cells/cubic mm) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  Platelets (1000 cells/cubic mm) -Day 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Platelets (1000 cells/cubic mm) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Platelets (1000 cells/cubic mm) -Day 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  Lymphocytes (1000 cells/cubic mm) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Lymphocytes (1000 cells/cubic mm) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  Lymphocytes (1000 cells/cubic mm) -Day 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Lymphocytes (1000 cells/cubic mm) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Lymphocytes (1000 cells/cubic mm) -Day 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 0/Enrollment: number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  Neutrophils (1000 cells/cubic mm) -Day 0/Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophils (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 15
  Neutrophils (1000 cells/cubic mm) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  Neutrophils (1000 cells/cubic mm) -Day 112 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 14
  Neutrophils (1000 cells/cubic mm) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophils (1000 cells/cubic mm) -Day 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  Neutrophils (1000 cells/cubic mm) -Day 280 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: The number (percentage) of participants with early discontinuation of vaccinations and reason for discontinuation was summarized by arm
Time Frame: Measured through Month 4
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
Participants
  Lost to Follow-Up | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
  Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Investigator reason | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Unsolicited AE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Solicited AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Did not discontinue SPA | 3 | 3 | 3 | 3 | 3 | 13 | 15 | 15 | 14 | 14

11. Primary Outcome: Number of Participants With Early Termination of Study and Reason for Early Termination
Description: The number (percentage) of participants with early termination of study and reason for early termination was summarized by arm
Time Frame: Measured through Month 6 in Part A and Month 10 in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
Participants
  Lost to Follow-Up | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
  Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Did not terminate Study | 3 | 3 | 3 | 3 | 3 | 13 | 16 | 16 | 16 | 14

12. Primary Outcome: Serum Concentration Levels of PGDM1400LS Among Participants Who Received All Scheduled Product Administrations
Description: Serum concentrations of PGDM1400LS at prespecified timepoints among participants who received all scheduled product administrations
Time Frame: Measured during Days 0, 0.0417 (1hr post 1st infusion), 3, 6, 28, 56, 112, 112.0417 (1hr post 2nd infusion)*, 168, 224*, and 280* Days with * are only available for T6-T10
Population: Overall Number of Participants Analyzed represents the number of enrolled participants. Number Analyzed- shows the number of participants with available data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
ug/ml
  PGDM1400LS - 0 | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.06] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04]
  PGDM1400LS - 0.0417 (Day 0 1 hr post-infusion): number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 14 | 15 | 16 | 16
  PGDM1400LS - 0.0417 (Day 0 1 hr post-infusion) | 96.49 [95.78 to 107.94] | 375.39 [348.03 to 385.94] | 1.19 [0.79 to 1.27] | 685.85 [673.75 to 708.24] | 2.92 [2.61 to 3.82] | 553.60 [514.21 to 689.08] | 6.38 [2.17 to 10.72] | 612.47 [545.95 to 662.88] | 11.36 [5.67 to 32.30] | 1190.49 [1107.99 to 1364.68]
  PGDM1400LS - 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 15 | 16
  PGDM1400LS - 3 | 95.69 [94.30 to 98.90] | 432.62 [404.40 to 467.57] | 146.40 [138.72 to 195.27] | 727.44 [699.95 to 753.49] | 447.90 [339.69 to 497.52] | 307.89 [274.47 to 336.27] | 141.12 [112.09 to 183.21] | 339.86 [298.13 to 379.21] | 212.99 [159.40 to 250.61] | 594.72 [537.59 to 760.35]
  PGDM1400LS - 6: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 14 | 16 | 16 | 16
  PGDM1400LS - 6 | 88.87 [83.00 to 89.43] | 361.09 [324.20 to 401.39] | 205.63 [181.88 to 244.03] | 603.62 [586.36 to 607.43] | 429.97 [343.03 to 508.78] | 266.18 [247.48 to 281.38] | 151.45 [129.36 to 209.50] | 265.27 [254.55 to 306.57] | 219.97 [168.17 to 274.74] | 499.59 [468.30 to 549.73]
  PGDM1400LS - 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 15 | 16 | 16 | 16
  PGDM1400LS - 28 | 69.81 [64.83 to 72.96] | 209.91 [206.92 to 265.82] | 140.04 [132.00 to 172.58] | 510.53 [490.21 to 532.83] | 313.98 [287.34 to 368.93] | 165.77 [154.51 to 192.02] | 113.85 [86.38 to 149.17] | 183.47 [177.72 to 186.74] | 154.89 [117.34 to 176.31] | 304.70 [281.78 to 364.51]
  PGDM1400LS - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 15 | 16 | 16 | 15
  PGDM1400LS - 56 | 43.02 [40.87 to 43.25] | 159.59 [149.70 to 171.80] | 97.86 [86.34 to 121.86] | 344.23 [325.91 to 366.04] | 214.17 [188.22 to 272.13] | 112.02 [102.31 to 127.35] | 75.03 [62.09 to 100.44] | 128.23 [109.13 to 137.01] | 102.92 [84.18 to 141.03] | 215.93 [182.69 to 257.77]
  PGDM1400LS - 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15 | 16 | 16 | 16 | 14
  PGDM1400LS - 112 | 19.24 [18.32 to 21.32] | 95.78 [89.48 to 104.45] | 50.75 [47.53 to 60.20] | 157.13 [155.26 to 166.78] | 105.81 [99.96 to 128.13] | 54.73 [48.45 to 67.89] | 42.29 [30.81 to 55.25] | 66.50 [53.14 to 76.49] | 46.32 [35.65 to 62.00] | 98.76 [82.29 to 128.24]
  PGDM1400LS - 112.0417 (Day 112 1 hr post-infusion): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 12 | 15 | 15 | 14 | 13
  PGDM1400LS - 112.0417 (Day 112 1 hr post-infusion) |  |  |  |  |  | 538.95 [405.11 to 606.24] | 55.77 [35.15 to 68.47] | 655.22 [598.31 to 755.91] | 63.50 [46.90 to 68.82] | 1347.38 [1120.57 to 1502.24]
  PGDM1400LS - 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 14 | 16 | 14 | 16 | 13
  PGDM1400LS - 168 | 9.26 [8.56 to 10.05] | 46.08 [41.34 to 49.57] | 19.19 [18.75 to 24.31] | 80.29 [72.14 to 94.05] | 46.78 [46.74 to 50.77] | 145.70 [117.67 to 152.43] | 120.50 [82.29 to 137.07] | 161.22 [132.14 to 169.46] | 123.02 [94.73 to 154.08] | 262.73 [231.67 to 311.74]
  PGDM1400LS - 224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 13
  PGDM1400LS - 224 |  |  |  |  |  | 62.34 [54.20 to 69.56] | 57.01 [39.58 to 68.37] | 71.55 [63.09 to 87.07] | 59.31 [44.62 to 75.73] | 124.27 [102.89 to 150.22]
  PGDM1400LS - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 16 | 14
  PGDM1400LS - 280 |  |  |  |  |  | 28.91 [26.39 to 34.65] | 23.87 [15.17 to 33.18] | 41.15 [32.14 to 44.20] | 32.96 [19.19 to 42.58] | 65.37 [50.14 to 72.40]

13. Primary Outcome: Serum Concentration Levels of PGT121.414LS Among Participants Who Received All Scheduled Product Administrations
Description: Serum concentrations of PGT121.414.LS at prespecified timepoints among participants who received all scheduled product administrations
Time Frame: Measured during Days 0, 0.0417 (1hr post 1st infusion), 3, 6, 28, 56, 112, 112.0417 (1hr post 2nd infusion), 168, 224, and 280
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ug/ml
  PGT121.414.LS - 0 | 0.10 [0.10 to 0.49] | 0.10 [0.10 to 0.10] | 0.10 [0.10 to 0.10] | 0.10 [0.10 to 0.10] | 0.10 [0.10 to 0.10]
  PGT121.414.LS - 0.0417 (Day 0 1 hr post-infusion): number analyzed (Participants) | 14 | 15 | 15 | 16 | 16
  PGT121.414.LS - 0.0417 (Day 0 1 hr post-infusion) | 903.30 [738.08 to 1176.36] | 4.97 [2.59 to 6.01] | 1021.49 [819.03 to 1158.71] | 7.22 [3.62 to 14.30] | 1875.25 [1518.96 to 2000.91]
  PGT121.414.LS - 3: number analyzed (Participants) | 16 | 15 | 16 | 15 | 16
  PGT121.414.LS - 3 | 386.38 [344.05 to 467.41] | 229.12 [149.99 to 249.87] | 431.97 [388.14 to 517.63] | 264.14 [210.82 to 308.86] | 679.23 [632.61 to 853.46]
  PGT121.414.LS - 6: number analyzed (Participants) | 15 | 14 | 16 | 16 | 16
  PGT121.414.LS - 6 | 336.42 [302.65 to 361.19] | 210.82 [166.11 to 257.88] | 348.90 [317.48 to 364.36] | 269.04 [239.84 to 302.81] | 623.84 [522.68 to 670.41]
  PGT121.414.LS - 28: number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
  PGT121.414.LS - 28 | 218.67 [196.79 to 232.36] | 155.20 [120.04 to 185.84] | 240.20 [230.27 to 247.46] | 199.02 [167.91 to 231.83] | 398.70 [371.81 to 520.71]
  PGT121.414.LS - 56: number analyzed (Participants) | 14 | 15 | 16 | 16 | 15
  PGT121.414.LS - 56 | 148.41 [138.80 to 175.11] | 104.16 [86.28 to 132.88] | 174.96 [155.05 to 191.54] | 144.98 [124.41 to 188.72] | 275.85 [241.89 to 345.03]
  PGT121.414.LS - 112: number analyzed (Participants) | 15 | 16 | 16 | 16 | 14
  PGT121.414.LS - 112 | 87.90 [69.71 to 102.35] | 58.88 [46.42 to 66.86] | 104.02 [73.83 to 118.95] | 72.58 [52.47 to 91.80] | 159.04 [129.42 to 190.73]
  PGT121.414.LS - 112.0417 (Day 112 1 hr post-infusion): number analyzed (Participants) | 12 | 15 | 15 | 14 | 13
  PGT121.414.LS - 112.0417 (Day 112 1 hr post-infusion) | 651.90 [537.81 to 809.14] | 72.48 [47.67 to 91.06] | 831.75 [760.79 to 888.09] | 80.52 [54.52 to 100.09] | 1759.82 [1585.83 to 1979.14]
  PGT121.414.LS - 168: number analyzed (Participants) | 14 | 16 | 14 | 16 | 13
  PGT121.414.LS - 168 | 188.24 [164.37 to 206.13] | 171.21 [108.50 to 194.51] | 235.47 [203.57 to 248.16] | 172.71 [128.87 to 207.83] | 386.92 [310.70 to 474.22]
  PGT121.414.LS - 224: number analyzed (Participants) | 13 | 16 | 16 | 16 | 13
  PGT121.414.LS - 224 | 104.50 [78.01 to 112.77] | 96.83 [54.28 to 102.47] | 120.60 [101.41 to 135.18] | 95.66 [62.73 to 126.24] | 217.87 [179.77 to 244.66]
  PGT121.414.LS - 280: number analyzed (Participants) | 13 | 16 | 16 | 16 | 14
  PGT121.414.LS - 280 | 55.87 [42.92 to 64.22] | 57.47 [34.73 to 64.47] | 75.78 [63.71 to 92.74] | 57.10 [28.27 to 80.37] | 111.83 [99.52 to 142.23]

14. Primary Outcome: Serum Concentration Levels of VRC07-523LS Among Participants Who Received All Scheduled Product Administrations
Description: Serum concentrations of VRC07-523LS at prespecified timepoints among participants who received all scheduled product administrations
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ug/ml
  VRC07-523LS - 0 | 0.02 [0.02 to 0.06] | 0.02 [0.02 to 0.03] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02]
  VRC07-523LS - 0.0417 (Day 0 1 hr post-infusion): number analyzed (Participants) | 14 | 14 | 15 | 16 | 16
  VRC07-523LS - 0.0417 (Day 0 1 hr post-infusion) | 663.07 [597.75 to 802.03] | 4.44 [2.53 to 5.30] | 695.08 [632.95 to 784.68] | 6.84 [4.48 to 10.38] | 1289.22 [1166.28 to 1462.65]
  VRC07-523LS - 3: number analyzed (Participants) | 16 | 15 | 16 | 15 | 16
  VRC07-523LS - 3 | 302.96 [266.68 to 362.20] | 129.45 [87.83 to 178.88] | 324.02 [280.57 to 349.53] | 188.96 [126.09 to 249.46] | 482.08 [435.83 to 610.29]
  VRC07-523LS - 6: number analyzed (Participants) | 15 | 14 | 16 | 16 | 16
  VRC07-523LS - 6 | 221.59 [205.34 to 245.54] | 129.81 [110.37 to 187.66] | 220.64 [210.89 to 237.89] | 191.63 [139.77 to 221.60] | 370.32 [328.89 to 447.89]
  VRC07-523LS - 28: number analyzed (Participants) | 16 | 15 | 16 | 16 | 16
  VRC07-523LS - 28 | 109.16 [92.54 to 122.88] | 75.29 [51.10 to 80.35] | 109.48 [97.32 to 124.65] | 98.05 [71.57 to 106.97] | 182.31 [158.46 to 210.75]
  VRC07-523LS - 56: number analyzed (Participants) | 14 | 15 | 16 | 16 | 15
  VRC07-523LS - 56 | 64.22 [54.59 to 71.72] | 41.90 [31.72 to 48.41] | 64.04 [60.04 to 78.78] | 58.30 [39.57 to 73.23] | 103.01 [92.30 to 116.08]
  VRC07-523LS - 112: number analyzed (Participants) | 15 | 16 | 16 | 16 | 14
  VRC07-523LS - 112 | 27.81 [24.59 to 37.18] | 17.58 [13.50 to 20.69] | 29.89 [22.43 to 39.49] | 21.99 [15.22 to 28.92] | 41.09 [34.66 to 58.76]
  VRC07-523LS - 112.0417 (Day 112 1 hr post-infusion): number analyzed (Participants) | 12 | 15 | 15 | 14 | 13
  VRC07-523LS - 112.0417 (Day 112 1 hr post-infusion) | 660.51 [511.46 to 796.07] | 22.38 [16.73 to 33.48] | 671.49 [578.23 to 761.13] | 29.32 [23.47 to 42.68] | 1344.90 [1149.85 to 1605.62]
  VRC07-523LS - 168: number analyzed (Participants) | 14 | 16 | 14 | 16 | 13
  VRC07-523LS - 168 | 74.16 [63.66 to 88.90] | 64.42 [40.86 to 74.97] | 81.72 [73.57 to 90.37] | 68.32 [51.44 to 86.28] | 124.88 [109.72 to 140.12]
  VRC07-523LS - 224: number analyzed (Participants) | 13 | 16 | 16 | 16 | 13
  VRC07-523LS - 224 | 31.52 [20.62 to 39.09] | 25.14 [17.75 to 31.48] | 31.16 [27.27 to 42.73] | 28.68 [18.01 to 37.42] | 42.35 [37.57 to 67.41]
  VRC07-523LS - 280: number analyzed (Participants) | 13 | 16 | 16 | 16 | 14
  VRC07-523LS - 280 | 11.32 [9.71 to 12.20] | 9.26 [7.16 to 12.18] | 12.84 [11.06 to 15.87] | 10.43 [5.51 to 20.38] | 17.33 [11.75 to 29.32]

15. Primary Outcome: Magnitude of Serum Neutralizing Activity (ie, Neutralizing Antibody Titers, Including ID50, ID80) for
Description: Magnitude of Serum Neutralizing Activity (ie, Neutralizing Antibody Titers, Including ID50, ID80) for Parts A and B
Time Frame: Measured during Days 0, 3, 6, 28, 56, 112, 168, 224*, and 280* Days with * are only available for T6-T10
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: titer
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
titer
  6540.v4.c1 - 50 - 0: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 9 | 9 | 10 | 10 | 9
  6540.v4.c1 - 50 - 0 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 150.00 [150.00 to 150.00] | 150.00 [150.00 to 150.00] | 150.00 [150.00 to 150.00] | 150.00 [150.00 to 150.00] | 150.00 [150.00 to 150.00]
  6540.v4.c1 - 50 - 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 9 | 9 | 10 | 10 | 9
  6540.v4.c1 - 50 - 3 | 18004.25 [16296.52 to 18714.19] | 86169.30 [72170.90 to 90818.29] | 37356.09 [33373.16 to 46693.84] | 210641.18 [176592.28 to 236319.49] | 104138.90 [82207.69 to 113630.00] | 78082.03 [60951.83 to 121013.02] | 38090.89 [26324.08 to 38905.20] | 94187.86 [76442.89 to 102587.67] | 44190.21 [38523.86 to 72645.07] | 155263.94 [145559.21 to 254422.80]
  6540.v4.c1 - 50 - 6: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 8 | 10 | 10 | 9
  6540.v4.c1 - 50 - 6 | 19536.62 [15684.20 to 19822.91] | 60315.19 [47368.30 to 60615.63] | 25318.17 [23065.01 to 32567.71] | 190567.11 [182226.74 to 211171.40] | 136086.26 [96705.97 to 173663.45] | 65735.36 [60026.66 to 80840.87] | 43426.88 [23192.42 to 60820.22] | 59253.58 [55517.03 to 75929.69] | 56244.87 [42079.23 to 67246.46] | 130118.65 [111524.54 to 175054.67]
  6540.v4.c1 - 50 - 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 9 | 10 | 9 | 8
  6540.v4.c1 - 50 - 28 | 11526.31 [9254.35 to 20291.81] | 35352.88 [33862.73 to 210041.52] | 20515.29 [17712.20 to 57337.84] | 95958.61 [85192.70 to 102149.48] | 228540.05 [132938.75 to 244799.10] | 32034.53 [29134.27 to 48227.96] | 23502.68 [19271.71 to 36751.52] | 46024.02 [31702.40 to 64639.69] | 40152.25 [31047.77 to 62268.95] | 63877.56 [60968.27 to 86642.55]
  6540.v4.c1 - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 8 | 10 | 9 | 8
  6540.v4.c1 - 50 - 56 | 3731.64 [3718.98 to 5700.14] | 32088.99 [25106.71 to 328424.34] | 18546.43 [14097.28 to 21778.94] | 35905.88 [29178.82 to 42702.50] | 48197.90 [31245.64 to 233644.78] | 17553.23 [15339.20 to 19304.85] | 10267.77 [8750.10 to 13263.23] | 17437.11 [13980.94 to 24584.85] | 15761.35 [10796.49 to 20269.17] | 31424.52 [21450.14 to 34972.42]
  6540.v4.c1 - 50 - 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 9 | 8 | 7
  6540.v4.c1 - 50 - 112 | 1294.45 [1075.53 to 1437.85] | 4856.32 [3780.45 to 6133.58] | 4108.53 [2842.06 to 4321.70] | 15403.44 [12837.51 to 24427.24] | 11323.91 [9460.00 to 11396.13] | 4452.10 [3725.43 to 5137.95] | 3652.50 [2112.79 to 4972.82] | 5287.92 [4595.94 to 8630.26] | 5614.97 [3629.30 to 9188.76] | 7748.86 [5045.92 to 13736.16]
  6540.v4.c1 - 50 - 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 7 | 8 | 6
  6540.v4.c1 - 50 - 168 | 633.13 [621.97 to 676.89] | 3477.51 [2384.10 to 3522.28] | 1055.97 [929.60 to 1226.42] | 3949.41 [3310.09 to 4618.12] | 1934.01 [1815.36 to 2030.59] | 22678.23 [18282.05 to 23955.40] | 18256.29 [9483.63 to 22053.37] | 21147.90 [19182.36 to 23969.75] | 21375.24 [19662.17 to 32268.48] | 40924.44 [35126.47 to 47267.91]
  6540.v4.c1 - 50 - 224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 8 | 8 | 8
  6540.v4.c1 - 50 - 224 |  |  |  |  |  | 7043.13 [5521.12 to 7712.26] | 4334.66 [2670.65 to 5512.28] | 6044.29 [5545.63 to 7605.48] | 5932.23 [5332.42 to 6993.82] | 12390.13 [11247.53 to 14418.62]
  6540.v4.c1 - 50 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 8 | 8 | 8
  6540.v4.c1 - 50 - 280 |  |  |  |  |  | 1948.28 [1795.74 to 2402.63] | 1744.59 [1508.26 to 2413.28] | 2578.49 [2011.20 to 2803.74] | 2679.28 [2216.32 to 4615.38] | 4869.88 [3888.36 to 5759.75]
  6540.v4.c1 - 80 - 0: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 9 | 9 | 10 | 10 | 9
  6540.v4.c1 - 80 - 0 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 150.00 [150.00 to 150.00] | 150.00 [150.00 to 150.00] | 150.00 [150.00 to 150.00] | 150.00 [150.00 to 150.00] | 150.00 [150.00 to 150.00]
  6540.v4.c1 - 80 - 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 9 | 9 | 10 | 10 | 9
  6540.v4.c1 - 80 - 3 | 4082.03 [3780.97 to 4265.98] | 18493.04 [15740.43 to 22035.52] | 6240.04 [5594.48 to 9338.30] | 38798.72 [36760.95 to 40611.61] | 16592.14 [13807.15 to 19986.46] | 23888.60 [17946.81 to 26204.21] | 8557.98 [6109.14 to 11696.77] | 20973.90 [19764.67 to 27220.65] | 10271.32 [7561.49 to 13069.24] | 42729.83 [32289.85 to 44389.46]
  6540.v4.c1 - 80 - 6: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 8 | 10 | 10 | 9
  6540.v4.c1 - 80 - 6 | 2890.20 [2784.12 to 3454.59] | 12699.51 [10238.51 to 13433.49] | 5965.47 [5170.04 to 8664.14] | 32217.59 [27030.31 to 32290.66] | 16526.64 [14367.75 to 21616.09] | 14844.38 [13397.01 to 20732.30] | 10843.79 [6389.07 to 14803.96] | 14559.28 [13221.35 to 18078.01] | 11285.60 [9943.26 to 15950.23] | 34219.06 [29156.53 to 49083.65]
  6540.v4.c1 - 80 - 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 9 | 10 | 9 | 8
  6540.v4.c1 - 80 - 28 | 1868.90 [1333.74 to 2335.96] | 5386.78 [4995.89 to 10173.70] | 3491.99 [2598.65 to 4133.99] | 14157.79 [13112.44 to 14741.65] | 10784.72 [9354.51 to 13264.06] | 7454.26 [6398.33 to 11592.09] | 6265.17 [3874.41 to 9890.65] | 10272.30 [7772.83 to 11426.41] | 11379.60 [7213.88 to 11735.73] | 15821.39 [12844.24 to 18105.67]
  6540.v4.c1 - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 8 | 10 | 9 | 8
  6540.v4.c1 - 80 - 56 | 746.39 [696.58 to 783.69] | 2718.94 [2711.53 to 2910.56] | 2672.84 [2221.22 to 2842.15] | 4626.30 [4091.12 to 4757.32] | 6475.97 [4503.69 to 7251.02] | 4039.11 [3949.73 to 5393.52] | 2175.54 [2055.93 to 3399.28] | 3958.18 [3111.29 to 4738.42] | 4572.76 [2837.10 to 5415.44] | 8098.32 [5523.62 to 9171.35]
  6540.v4.c1 - 80 - 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 9 | 8 | 7
  6540.v4.c1 - 80 - 112 | 192.85 [186.48 to 276.98] | 826.94 [685.28 to 940.14] | 437.47 [406.28 to 632.04] | 2065.96 [1913.21 to 3264.76] | 1283.49 [1157.58 to 1922.85] | 1384.65 [979.44 to 1459.86] | 754.64 [567.02 to 1262.59] | 1179.07 [904.10 to 1858.06] | 1245.31 [808.02 to 2033.39] | 1425.73 [1235.60 to 3642.00]
  6540.v4.c1 - 80 - 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 7 | 8 | 6
  6540.v4.c1 - 80 - 168 | 24.02 [14.51 to 26.64] | 492.93 [364.62 to 575.80] | 183.14 [176.99 to 212.84] | 493.97 [438.70 to 827.81] | 442.94 [395.34 to 478.23] | 6030.57 [5008.24 to 6270.58] | 4132.63 [2366.80 to 5047.10] | 4763.95 [4601.31 to 6325.77] | 5709.83 [4855.07 to 7392.76] | 8816.20 [8355.48 to 9975.19]
  6540.v4.c1 - 80 - 224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 8 | 8 | 8
  6540.v4.c1 - 80 - 224 |  |  |  |  |  | 1492.16 [1274.73 to 1529.01] | 890.67 [628.01 to 964.92] | 1536.64 [1388.43 to 1800.76] | 1375.26 [1227.32 to 1629.20] | 2624.72 [2289.68 to 2875.02]
  6540.v4.c1 - 80 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 8 | 8 | 8
  6540.v4.c1 - 80 - 280 |  |  |  |  |  | 504.34 [460.99 to 576.34] | 468.48 [398.69 to 553.73] | 626.33 [450.05 to 716.94] | 620.44 [479.35 to 995.12] | 957.91 [782.20 to 1124.43]
  CH505TF.N334S.N160A.N280D.1 - 50 - 0: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 9 | 9 | 10 | 10 | 9
  CH505TF.N334S.N160A.N280D.1 - 50 - 0 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 150.00 [5.00 to 150.00] | 150.00 [150.00 to 150.00] | 150.00 [41.25 to 150.00] | 150.00 [5.00 to 150.00] | 150.00 [150.00 to 150.00]
  CH505TF.N334S.N160A.N280D.1 - 50 - 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 9 | 9 | 10 | 10 | 9
  CH505TF.N334S.N160A.N280D.1 - 50 - 3 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 111359.04 [92054.13 to 174231.52] | 31531.64 [22933.66 to 41518.28] | 101622.05 [65815.14 to 155208.76] | 42738.95 [35264.24 to 80896.35] | 174911.25 [145783.28 to 268899.36]
  CH505TF.N334S.N160A.N280D.1 - 50 - 6: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 8 | 10 | 10 | 9
  CH505TF.N334S.N160A.N280D.1 - 50 - 6 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 76729.85 [67368.47 to 89654.37] | 53408.16 [37946.27 to 62285.80] | 63097.95 [59894.01 to 126480.51] | 63289.84 [42740.43 to 76527.82] | 114514.34 [97655.90 to 187033.29]
  CH505TF.N334S.N160A.N280D.1 - 50 - 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 9 | 10 | 9 | 8
  CH505TF.N334S.N160A.N280D.1 - 50 - 28 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 42765.16 [24583.81 to 60909.27] | 29399.28 [22355.27 to 37150.95] | 43229.29 [31019.30 to 56172.37] | 44216.61 [35731.35 to 50090.90] | 75530.56 [67863.44 to 90113.66]
  CH505TF.N334S.N160A.N280D.1 - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 8 | 10 | 9 | 8
  CH505TF.N334S.N160A.N280D.1 - 50 - 56 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 26446.02 [20358.58 to 34208.79] | 15139.18 [12628.24 to 17021.59] | 26799.63 [20592.70 to 38198.19] | 20066.68 [17046.16 to 26833.93] | 58752.83 [32646.43 to 79415.94]
  CH505TF.N334S.N160A.N280D.1 - 50 - 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 9 | 8 | 7
  CH505TF.N334S.N160A.N280D.1 - 50 - 112 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 12.63 [8.81 to 13.61] | 5.00 [5.00 to 8.04] | 9790.75 [7723.35 to 11072.58] | 8621.43 [4924.97 to 11629.46] | 12309.30 [8580.90 to 16389.17] | 10878.05 [6001.01 to 21303.79] | 23825.19 [15108.51 to 28662.83]
  CH505TF.N334S.N160A.N280D.1 - 50 - 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 7 | 8 | 6
  CH505TF.N334S.N160A.N280D.1 - 50 - 168 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 11.35 [10.93 to 11.55] | 5.00 [5.00 to 11.16] | 36402.30 [29858.83 to 36428.19] | 40368.23 [29784.33 to 47492.89] | 39562.48 [27812.93 to 49942.15] | 36565.68 [31725.14 to 52573.96] | 88221.37 [81072.30 to 109631.90]
  CH505TF.N334S.N160A.N280D.1 - 50 - 224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 8 | 8 | 8
  CH505TF.N334S.N160A.N280D.1 - 50 - 224 |  |  |  |  |  | 19975.51 [13481.68 to 21054.36] | 12846.42 [8262.33 to 15054.90] | 21710.66 [16086.53 to 24826.44] | 19689.54 [12874.10 to 22199.23] | 37227.47 [36036.61 to 44972.22]
  CH505TF.N334S.N160A.N280D.1 - 50 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 8 | 8 | 8
  CH505TF.N334S.N160A.N280D.1 - 50 - 280 |  |  |  |  |  | 6386.89 [6059.01 to 7838.87] | 7614.93 [5751.88 to 9392.22] | 10111.45 [8816.90 to 11593.81] | 11651.39 [6453.99 to 17367.78] | 15470.09 [13140.16 to 26177.69]
  CH505TF.N334S.N160A.N280D.1 - 80 - 0: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 9 | 9 | 10 | 10 | 9
  CH505TF.N334S.N160A.N280D.1 - 80 - 0 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 150.00 [5.00 to 150.00] | 150.00 [150.00 to 150.00] | 150.00 [41.25 to 150.00] | 150.00 [41.25 to 150.00] | 150.00 [150.00 to 150.00]
  CH505TF.N334S.N160A.N280D.1 - 80 - 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 9 | 9 | 10 | 10 | 9
  CH505TF.N334S.N160A.N280D.1 - 80 - 3 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 39720.65 [25883.40 to 54402.57] | 12451.16 [10170.48 to 15957.46] | 30936.66 [23216.20 to 59865.17] | 13229.33 [11411.01 to 21676.60] | 56218.55 [38214.75 to 81900.83]
  CH505TF.N334S.N160A.N280D.1 - 80 - 6: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 8 | 10 | 10 | 9
  CH505TF.N334S.N160A.N280D.1 - 80 - 6 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 23276.79 [19493.60 to 28243.02] | 14051.96 [11299.73 to 16681.05] | 22619.87 [18319.07 to 39552.68] | 18368.24 [12960.45 to 26431.58] | 36881.20 [29376.52 to 53533.46]
  CH505TF.N334S.N160A.N280D.1 - 80 - 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 9 | 10 | 9 | 8
  CH505TF.N334S.N160A.N280D.1 - 80 - 28 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 11808.90 [8701.84 to 17426.27] | 11401.34 [7795.13 to 13566.30] | 16750.64 [9477.15 to 17986.88] | 15171.56 [11153.22 to 16016.70] | 22791.38 [20499.22 to 31307.64]
  CH505TF.N334S.N160A.N280D.1 - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 8 | 10 | 9 | 8
  CH505TF.N334S.N160A.N280D.1 - 80 - 56 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 9310.84 [7458.89 to 12333.71] | 5301.73 [4489.83 to 5820.16] | 10545.50 [7477.06 to 13598.23] | 5803.64 [5477.07 to 9610.62] | 18420.21 [14420.38 to 22793.06]
  CH505TF.N334S.N160A.N280D.1 - 80 - 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 9 | 8 | 7
  CH505TF.N334S.N160A.N280D.1 - 80 - 112 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 3115.33 [2633.93 to 4133.73] | 2222.96 [1775.74 to 4060.71] | 4217.73 [2659.19 to 5629.76] | 3491.96 [2380.38 to 6432.59] | 6910.25 [4918.82 to 9930.57]
  CH505TF.N334S.N160A.N280D.1 - 80 - 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 7 | 8 | 6
  CH505TF.N334S.N160A.N280D.1 - 80 - 168 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 14050.60 [13619.78 to 14086.03] | 13435.34 [8391.38 to 16451.07] | 13643.32 [11034.37 to 16974.48] | 12171.52 [10663.22 to 14135.50] | 29423.14 [24552.36 to 29831.69]
  CH505TF.N334S.N160A.N280D.1 - 80 - 224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 8 | 8 | 8
  CH505TF.N334S.N160A.N280D.1 - 80 - 224 |  |  |  |  |  | 5670.50 [4203.45 to 6305.68] | 4087.73 [3157.60 to 5263.09] | 6640.69 [5430.59 to 8694.89] | 7348.03 [4254.03 to 8059.42] | 13020.14 [11544.71 to 14707.77]
  CH505TF.N334S.N160A.N280D.1 - 80 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 8 | 8 | 8
  CH505TF.N334S.N160A.N280D.1 - 80 - 280 |  |  |  |  |  | 2210.13 [1794.48 to 2311.82] | 2308.80 [1820.20 to 3199.86] | 3869.87 [3306.85 to 4252.37] | 4586.73 [2657.94 to 5574.31] | 5429.12 [4566.64 to 7689.83]
  CNE55.N160K - 50 - 0: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 9 | 10 | 10 | 10 | 10
  CNE55.N160K - 50 - 0 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  CNE55.N160K - 50 - 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 9 | 10 | 11 | 10 | 10
  CNE55.N160K - 50 - 3 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5724.38 [2998.04 to 6742.43] | 1454.65 [987.44 to 1883.54] | 3654.32 [3549.50 to 4492.37] | 2816.67 [1877.01 to 5026.68] | 7184.43 [5402.77 to 9699.20]
  CNE55.N160K - 50 - 6: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 9 | 10 | 10 | 10
  CNE55.N160K - 50 - 6 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 2036.61 [1502.85 to 2518.73] | 882.99 [785.07 to 1531.96] | 2376.08 [1770.84 to 3485.61] | 3008.78 [1402.43 to 5193.25] | 5362.34 [3440.08 to 6842.72]
  CNE55.N160K - 50 - 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 9 | 10 | 10 | 10 | 10
  CNE55.N160K - 50 - 28 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 690.34 [627.11 to 2405.47] | 512.34 [470.85 to 694.57] | 1071.55 [1024.20 to 1467.32] | 1138.94 [426.97 to 1388.66] | 1692.69 [1361.81 to 2219.53]
  CNE55.N160K - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 8 | 10 | 9 | 8
  CNE55.N160K - 50 - 56 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 712.10 [437.32 to 1188.64] | 330.68 [204.09 to 451.92] | 733.53 [629.29 to 902.64] | 465.56 [411.48 to 672.54] | 1173.82 [857.74 to 1451.62]
  CNE55.N160K - 50 - 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 9 | 8 | 7
  CNE55.N160K - 50 - 112 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 142.06 [128.69 to 209.17] | 82.83 [77.40 to 90.45] | 216.97 [113.83 to 277.82] | 277.60 [123.67 to 505.04] | 564.30 [318.38 to 700.87]
  CNE55.N160K - 50 - 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 7 | 8 | 6
  CNE55.N160K - 50 - 168 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 12.24] | 13.95 [9.47 to 14.01] | 580.36 [348.99 to 648.33] | 452.05 [270.81 to 691.32] | 398.50 [376.88 to 598.77] | 395.85 [249.97 to 596.12] | 803.11 [623.97 to 836.58]
  CNE55.N160K - 50 - 224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 9 | 8 | 8
  CNE55.N160K - 50 - 224 |  |  |  |  |  | 112.82 [91.56 to 153.43] | 145.43 [76.98 to 202.42] | 123.78 [110.59 to 251.40] | 262.75 [140.25 to 387.68] | 277.69 [183.23 to 565.76]
  CNE55.N160K - 50 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 8 | 9 | 9
  CNE55.N160K - 50 - 280 |  |  |  |  |  | 47.06 [41.59 to 49.03] | 45.88 [34.13 to 61.55] | 67.95 [47.76 to 112.81] | 59.54 [28.72 to 87.74] | 130.02 [86.39 to 141.12]
  CNE55.N160K - 80 - 0: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 9 | 10 | 10 | 10 | 10
  CNE55.N160K - 80 - 0 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  CNE55.N160K - 80 - 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 9 | 10 | 11 | 10 | 10
  CNE55.N160K - 80 - 3 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 728.14 [589.60 to 946.91] | 171.01 [143.12 to 288.02] | 623.34 [596.54 to 763.48] | 341.19 [233.12 to 431.25] | 1590.53 [1283.27 to 1755.00]
  CNE55.N160K - 80 - 6: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 9 | 10 | 10 | 10
  CNE55.N160K - 80 - 6 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 321.65 [272.40 to 397.22] | 150.73 [121.58 to 339.99] | 483.85 [355.86 to 530.10] | 344.46 [200.75 to 488.87] | 881.45 [728.12 to 960.47]
  CNE55.N160K - 80 - 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 9 | 10 | 10 | 10 | 10
  CNE55.N160K - 80 - 28 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 179.90 [170.46 to 213.35] | 81.67 [42.26 to 101.45] | 207.57 [136.87 to 282.30] | 125.74 [82.92 to 188.61] | 352.64 [308.74 to 458.91]
  CNE55.N160K - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 8 | 10 | 9 | 8
  CNE55.N160K - 80 - 56 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 75.92 [62.83 to 145.79] | 29.74 [26.05 to 53.11] | 101.47 [72.92 to 123.23] | 76.61 [42.93 to 115.27] | 162.81 [143.03 to 172.93]
  CNE55.N160K - 80 - 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 9 | 8 | 7
  CNE55.N160K - 80 - 112 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 17.74 [6.30 to 37.49] | 23.96 [18.12 to 27.87] | 27.53 [25.92 to 53.40] | 31.34 [22.25 to 37.02] | 55.81 [27.29 to 60.05]
  CNE55.N160K - 80 - 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 8 | 7 | 8 | 6
  CNE55.N160K - 80 - 168 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 84.51 [59.66 to 85.65] | 59.59 [48.22 to 72.27] | 74.82 [64.99 to 108.97] | 64.31 [44.73 to 82.40] | 103.93 [81.38 to 113.65]
  CNE55.N160K - 80 - 224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 8 | 9 | 8 | 8
  CNE55.N160K - 80 - 224 |  |  |  |  |  | 24.20 [22.44 to 32.11] | 18.20 [14.24 to 25.21] | 39.01 [33.56 to 49.50] | 28.50 [20.84 to 44.34] | 43.58 [34.61 to 66.82]
  CNE55.N160K - 80 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 8 | 9 | 9
  CNE55.N160K - 80 - 280 |  |  |  |  |  | 22.66 [19.63 to 28.22] | 15.08 [13.42 to 19.11] | 18.48 [16.03 to 23.03] | 17.11 [5.00 to 21.63] | 23.39 [20.32 to 24.47]

16. Primary Outcome: Magnitude Breadth of Serum Neutralizing Activity (ie, Neutralizing Antibody Titers, Including ID50, ID80) for Parts A and B
Description: Magnitude breadth of neutralizing activity measured with Env pseudotyped viruses specific for either PGDM1400LS, VRC07-523LS or PGT121.414LS in TZM-bl cells at prespecified timepoints among participants who received all scheduled product administrations for Parts A and B.
Time Frame: Measured during Days 56 and 168* Days with * are only available for T6-T10
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: log10(titer)
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
log10(titer)
  50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  50 - 56 | 1.83 [1.82 to 1.88] | 2.35 [2.34 to 2.36] | 2.19 [2.09 to 2.19] | 2.33 [2.31 to 2.35] | 2.26 [2.26 to 2.39] | 4.24 [4.20 to 4.34] | 3.97 [3.90 to 4.04] | 4.22 [4.14 to 4.30] | 4.06 [3.99 to 4.29] | 4.50 [4.43 to 4.61]
  50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  50 - 168 |  |  |  |  |  | 4.17 [4.06 to 4.28] | 4.07 [3.94 to 4.15] | 4.36 [4.31 to 4.40] | 4.17 [3.91 to 4.28] | 4.42 [4.40 to 4.68]
  80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  80 - 56 | 1.42 [1.42 to 1.47] | 1.76 [1.74 to 1.78] | 1.60 [1.53 to 1.67] | 1.77 [1.76 to 1.78] | 1.81 [1.73 to 1.86] | 3.62 [3.57 to 3.72] | 3.40 [3.31 to 3.51] | 3.69 [3.59 to 3.72] | 3.49 [3.36 to 3.63] | 3.92 [3.85 to 3.98]
  80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  80 - 168 |  |  |  |  |  | 3.57 [3.42 to 3.70] | 3.41 [3.31 to 3.57] | 3.71 [3.63 to 3.75] | 3.54 [3.34 to 3.67] | 3.87 [3.84 to 4.05]

17. Secondary Outcome: Magnitude of Neutralizing Activity Against Env-pseudotyped Viruses in TZM-bl Cells for Part A and B and Clinical Product Assayed at Same Time.
Description: Magnitude of neutralizing activity against a panel of Env-pseudotyped reference viruses that are sensitive to all three bnAbs in TZM-bl cells at selected timepoints for all participants in all groups regardless of how many product administrations and how much product they received
Time Frame: Day 56 and Day 168* corresponding to Month 2 and Month 6* of the study. Days with * are only available for T6-T10
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: titer
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
titer
  H703_0472_030s - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H703_0472_030s - 50 - 56 | 10.00 [10.00 to 10.00] | 133.29 [132.09 to 191.11] | 10.00 [10.00 to 151.06] | 10.00 [10.00 to 10.00] | 48.80 [29.40 to 391.07] | 28867.34 [20743.95 to 39580.10] | 9124.56 [7448.63 to 12654.71] | 19418.37 [15353.70 to 26741.45] | 13043.79 [8991.62 to 20691.21] | 29487.53 [20734.74 to 36956.15]
  H703_0472_030s - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H703_0472_030s - 50 - 168 |  |  |  |  |  | 15360.16 [13131.22 to 18028.60] | 10917.47 [8209.55 to 12007.01] | 18239.03 [13007.53 to 21793.19] | 11090.80 [7072.91 to 17886.50] | 20497.50 [17559.38 to 26140.18]
  H703_0472_030s - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H703_0472_030s - 80 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 9199.85 [6368.56 to 9834.28] | 2649.77 [2481.71 to 4100.21] | 6707.18 [4557.14 to 8128.45] | 4266.58 [2497.77 to 7337.54] | 9751.86 [6866.64 to 12886.76]
  H703_0472_030s - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H703_0472_030s - 80 - 168 |  |  |  |  |  | 4947.38 [4807.10 to 5843.26] | 3553.36 [2820.22 to 4158.40] | 5255.50 [4585.44 to 8058.00] | 3885.02 [2367.69 to 5345.99] | 8034.77 [7410.92 to 9130.71]
  H703_2117_110_RE_e2A10s - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H703_2117_110_RE_e2A10s - 50 - 56 | 44472.66 [29406.06 to 46797.85] | 170780.42 [122746.39 to 173544.27] | 41897.36 [36512.97 to 76003.51] | 107823.15 [104194.71 to 111675.54] | 77124.52 [64268.48 to 78146.68] | 168357.12 [100766.88 to 196927.70] | 66253.95 [60899.93 to 82832.43] | 107878.92 [70813.58 to 137241.39] | 102278.55 [75056.44 to 114569.94] | 256420.14 [203041.94 to 545729.61]
  H703_2117_110_RE_e2A10s - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H703_2117_110_RE_e2A10s - 50 - 168 |  |  |  |  |  | 86881.47 [78522.12 to 90414.47] | 71999.91 [43000.38 to 81379.06] | 132113.38 [112056.82 to 163289.85] | 81157.57 [52587.55 to 139949.62] | 148145.98 [127852.90 to 1209608.52]
  H703_2117_110_RE_e2A10s - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H703_2117_110_RE_e2A10s - 80 - 56 | 7831.73 [6782.93 to 8475.95] | 42634.56 [36579.79 to 44503.08] | 13815.72 [12398.39 to 21192.79] | 29824.76 [28415.28 to 29956.70] | 19004.67 [16573.19 to 21171.18] | 41391.40 [31015.41 to 42404.04] | 21151.88 [17098.51 to 24883.17] | 33571.08 [29386.77 to 47067.16] | 28888.77 [18829.88 to 46316.27] | 64290.02 [49632.03 to 107726.55]
  H703_2117_110_RE_e2A10s - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H703_2117_110_RE_e2A10s - 80 - 168 |  |  |  |  |  | 28897.55 [25500.79 to 31831.18] | 23002.49 [16945.94 to 31779.52] | 39488.60 [37566.74 to 40215.25] | 26000.40 [20112.19 to 33882.23] | 58317.53 [44928.83 to 130565.38]
  H703_2304_150_RE_cs - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H703_2304_150_RE_cs - 50 - 56 | 1208.31 [1190.68 to 1327.46] | 7065.76 [6006.06 to 7167.62] | 3238.87 [2524.67 to 3867.71] | 5823.93 [5125.95 to 7568.17] | 8454.64 [5854.08 to 13182.48] | 33327.66 [29725.61 to 89182.04] | 19116.20 [14812.53 to 27698.26] | 29807.82 [21350.86 to 39150.71] | 23789.32 [18834.67 to 42987.41] | 57599.35 [41356.47 to 110040.00]
  H703_2304_150_RE_cs - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H703_2304_150_RE_cs - 50 - 168 |  |  |  |  |  | 23924.35 [19423.14 to 40216.80] | 15632.62 [13448.63 to 22284.53] | 26314.31 [24931.64 to 33052.24] | 16910.80 [11004.20 to 25598.01] | 39775.62 [26215.22 to 47397.58]
  H703_2304_150_RE_cs - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H703_2304_150_RE_cs - 80 - 56 | 10.00 [10.00 to 44.69] | 141.31 [140.79 to 220.81] | 126.83 [68.41 to 128.15] | 10.00 [10.00 to 10.00] | 120.68 [65.34 to 324.43] | 10157.60 [6278.87 to 11793.02] | 5333.96 [3559.08 to 6638.95] | 8684.03 [5706.35 to 10290.43] | 5054.29 [3918.81 to 9293.38] | 15033.13 [9364.53 to 23332.90]
  H703_2304_150_RE_cs - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H703_2304_150_RE_cs - 80 - 168 |  |  |  |  |  | 5888.07 [4796.79 to 8184.63] | 4043.14 [3259.53 to 5743.73] | 6921.19 [6026.46 to 9194.93] | 5397.31 [3636.99 to 7495.72] | 9955.22 [9218.46 to 13984.86]
  H703_2805_080Es - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H703_2805_080Es - 50 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 6702.06 [5866.82 to 9301.05] | 3827.22 [2613.18 to 4515.86] | 7284.91 [5625.40 to 8149.53] | 5429.73 [2748.64 to 8202.83] | 11642.31 [10249.54 to 13495.04]
  H703_2805_080Es - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H703_2805_080Es - 50 - 168 |  |  |  |  |  | 8055.72 [7407.58 to 8275.73] | 4998.26 [2925.21 to 6797.41] | 8771.74 [6855.85 to 12328.36] | 5430.58 [2646.49 to 10889.28] | 14806.94 [14317.38 to 17968.28]
  H703_2805_080Es - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H703_2805_080Es - 80 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 1550.43 [1368.54 to 1955.72] | 844.66 [627.56 to 989.87] | 1720.99 [1297.38 to 1997.91] | 1147.58 [604.60 to 1901.81] | 2766.88 [2166.58 to 3882.55]
  H703_2805_080Es - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H703_2805_080Es - 80 - 168 |  |  |  |  |  | 1681.16 [1421.99 to 2164.35] | 995.89 [824.91 to 1326.43] | 1882.14 [1081.20 to 2409.03] | 1683.91 [797.11 to 2371.55] | 3200.56 [2846.06 to 3408.02]
  H704_0128_220_RE_pb001_s - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_0128_220_RE_pb001_s - 50 - 56 | 2054.33 [2003.30 to 2169.36] | 8993.79 [8560.45 to 9703.10] | 3980.77 [3969.29 to 6453.81] | 18366.52 [16650.38 to 20584.03] | 11331.69 [9614.73 to 11934.66] | 39127.87 [29796.73 to 56970.43] | 22594.30 [18778.06 to 31045.85] | 39373.01 [30382.05 to 60718.47] | 45781.87 [31494.28 to 65215.52] | 80954.57 [60919.34 to 112568.94]
  H704_0128_220_RE_pb001_s - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_0128_220_RE_pb001_s - 50 - 168 |  |  |  |  |  | 45487.53 [32930.99 to 52015.30] | 31670.23 [21910.04 to 38112.08] | 49696.36 [47116.69 to 61935.77] | 33050.62 [22841.22 to 44745.34] | 77026.80 [57622.62 to 82921.82]
  H704_0128_220_RE_pb001_s - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_0128_220_RE_pb001_s - 80 - 56 | 639.49 [604.61 to 660.92] | 3051.10 [2940.96 to 3347.66] | 1349.82 [1218.83 to 1942.00] | 5744.76 [5525.98 to 6284.43] | 5206.67 [4037.48 to 5315.05] | 10658.64 [8477.88 to 12474.23] | 6686.16 [5025.48 to 8240.72] | 11570.84 [9389.13 to 14516.57] | 10688.77 [6119.35 to 17534.53] | 20826.12 [18873.78 to 30079.57]
  H704_0128_220_RE_pb001_s - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_0128_220_RE_pb001_s - 80 - 168 |  |  |  |  |  | 9737.36 [8355.11 to 13038.30] | 8441.28 [5095.94 to 10008.53] | 14323.05 [14107.54 to 14602.08] | 8126.62 [4361.08 to 10869.81] | 20457.55 [18349.90 to 28056.34]
  H704_0445_180_RE_con_s - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_0445_180_RE_con_s - 50 - 56 | 42.32 [40.58 to 48.76] | 147.95 [147.00 to 155.33] | 82.59 [74.56 to 98.71] | 278.40 [272.15 to 287.49] | 267.65 [217.90 to 300.79] | 1238.90 [899.90 to 1365.14] | 543.16 [504.13 to 708.99] | 1061.53 [945.13 to 1237.50] | 921.85 [573.52 to 1091.16] | 1798.57 [1367.90 to 2022.31]
  H704_0445_180_RE_con_s - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_0445_180_RE_con_s - 50 - 168 |  |  |  |  |  | 1047.87 [838.46 to 1222.54] | 837.65 [514.52 to 930.68] | 1120.53 [883.26 to 1404.03] | 867.36 [477.86 to 1100.31] | 1932.03 [1806.40 to 2650.67]
  H704_0445_180_RE_con_s - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_0445_180_RE_con_s - 80 - 56 | 10.00 [10.00 to 10.00] | 49.04 [47.60 to 50.33] | 20.64 [15.32 to 28.33] | 88.96 [84.17 to 95.94] | 70.41 [61.04 to 78.91] | 357.98 [274.26 to 409.14] | 176.65 [164.67 to 236.61] | 365.00 [308.22 to 404.53] | 300.98 [190.35 to 347.92] | 488.52 [413.64 to 674.45]
  H704_0445_180_RE_con_s - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_0445_180_RE_con_s - 80 - 168 |  |  |  |  |  | 322.12 [265.83 to 363.06] | 252.05 [179.13 to 286.69] | 316.37 [291.65 to 390.11] | 287.66 [177.14 to 372.87] | 581.13 [538.99 to 659.41]
  H704_0855_080_EsN - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_0855_080_EsN - 50 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 16066.82 [14056.31 to 18402.66] | 8998.09 [7166.75 to 13034.63] | 17822.44 [14363.41 to 23859.96] | 14887.80 [9984.72 to 22224.24] | 32917.33 [25943.41 to 44162.82]
  H704_0855_080_EsN - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_0855_080_EsN - 50 - 168 |  |  |  |  |  | 22218.02 [17371.37 to 25701.41] | 17928.86 [12155.92 to 27828.30] | 54853.25 [15500.39 to 58327.93] | 18946.53 [14197.96 to 29900.68] | 33836.22 [20677.29 to 53724.66]
  H704_0855_080_EsN - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_0855_080_EsN - 80 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 4007.12 [3657.42 to 4586.10] | 1816.41 [1583.17 to 2498.04] | 4663.11 [3704.39 to 5220.77] | 2628.16 [1661.81 to 4970.95] | 7924.07 [5528.17 to 11016.89]
  H704_0855_080_EsN - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_0855_080_EsN - 80 - 168 |  |  |  |  |  | 3730.92 [3175.84 to 5717.46] | 2646.71 [1857.93 to 3914.69] | 4616.80 [3601.84 to 8276.70] | 2649.60 [1277.53 to 4680.81] | 5920.02 [5246.91 to 8247.29]
  H704_0907_130sN - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_0907_130sN - 50 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 40369.74 [33405.71 to 51442.82] | 24700.41 [16859.64 to 29059.94] | 40507.06 [27692.80 to 58739.96] | 23847.08 [20555.60 to 48305.50] | 76855.39 [49863.71 to 106651.34]
  H704_0907_130sN - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_0907_130sN - 50 - 168 |  |  |  |  |  | 31018.25 [28416.50 to 37206.64] | 33646.19 [23296.90 to 42967.90] | 46842.83 [40163.41 to 50937.11] | 27190.76 [20791.79 to 54818.19] | 85799.88 [79542.43 to 157961.18]
  H704_0907_130sN - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_0907_130sN - 80 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 11734.09 [9715.46 to 13570.48] | 8733.83 [6040.65 to 10087.01] | 13241.02 [9901.32 to 17689.99] | 7957.70 [6355.60 to 13878.02] | 24924.38 [22576.48 to 28079.32]
  H704_0907_130sN - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_0907_130sN - 80 - 168 |  |  |  |  |  | 10566.71 [9337.60 to 12113.74] | 11294.94 [8173.07 to 12895.74] | 12934.70 [12590.47 to 14107.93] | 10396.23 [8686.59 to 16761.83] | 31529.07 [26401.86 to 36070.90]
  H704_1180_070EsN - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_1180_070EsN - 50 - 56 | 52.48 [41.62 to 65.44] | 479.06 [437.20 to 504.66] | 264.99 [174.37 to 315.37] | 796.76 [640.43 to 914.98] | 481.05 [394.15 to 663.23] | 2124.99 [1635.18 to 2432.53] | 755.24 [681.67 to 1107.32] | 1688.12 [1219.06 to 2025.41] | 1368.86 [967.52 to 2020.95] | 2690.94 [1796.42 to 3132.60]
  H704_1180_070EsN - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_1180_070EsN - 50 - 168 |  |  |  |  |  | 1698.60 [1337.49 to 1841.09] | 1328.75 [1025.40 to 1958.07] | 2019.75 [1740.66 to 4478.74] | 1448.31 [677.06 to 2041.07] | 2596.69 [1798.41 to 3678.49]
  H704_1180_070EsN - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_1180_070EsN - 80 - 56 | 10.00 [10.00 to 10.00] | 21.85 [15.92 to 41.97] | 10.00 [10.00 to 22.71] | 79.78 [70.96 to 86.48] | 84.29 [69.94 to 96.60] | 291.52 [268.66 to 345.28] | 157.57 [136.86 to 225.98] | 330.84 [281.90 to 419.48] | 157.47 [135.15 to 361.39] | 416.93 [369.52 to 675.25]
  H704_1180_070EsN - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_1180_070EsN - 80 - 168 |  |  |  |  |  | 253.39 [149.75 to 335.90] | 218.16 [139.95 to 302.97] | 348.17 [201.95 to 395.01] | 245.61 [152.22 to 348.20] | 399.61 [343.40 to 480.31]
  H704_1528_240_RE_pblib_001_s - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_1528_240_RE_pblib_001_s - 50 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 36426.42 [34043.50 to 55625.24] | 23445.12 [17608.38 to 28520.47] | 50167.98 [21797.78 to 78616.61] | 27489.85 [19627.80 to 41960.91] | 106157.59 [71385.41 to 142954.07]
  H704_1528_240_RE_pblib_001_s - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_1528_240_RE_pblib_001_s - 50 - 168 |  |  |  |  |  | 38260.68 [17684.51 to 43129.21] | 22333.24 [11198.84 to 29278.06] | 61237.42 [46009.12 to 127217.07] | 22870.26 [12696.10 to 40185.65] | 108220.51 [58749.69 to 168168.59]
  H704_1528_240_RE_pblib_001_s - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_1528_240_RE_pblib_001_s - 80 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 11959.12 [10432.91 to 14039.98] | 6762.32 [5403.51 to 9386.48] | 15756.62 [6676.25 to 18379.60] | 7703.47 [6423.19 to 9241.14] | 29557.51 [19574.58 to 36531.86]
  H704_1528_240_RE_pblib_001_s - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_1528_240_RE_pblib_001_s - 80 - 168 |  |  |  |  |  | 10865.19 [3217.66 to 12999.99] | 7091.64 [3178.85 to 9617.96] | 16773.85 [13168.14 to 18620.83] | 7753.47 [3915.85 to 13653.99] | 29248.76 [16641.20 to 38732.32]
  H704_1535_030sN - 50 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_1535_030sN - 50 - 56 | 10.00 [10.00 to 15.57] | 73.40 [65.48 to 83.40] | 53.90 [48.68 to 61.44] | 163.91 [145.08 to 164.93] | 121.63 [115.95 to 123.87] | 18072.17 [14792.44 to 20837.51] | 12696.91 [9827.76 to 19332.55] | 23023.75 [16462.06 to 31406.05] | 17665.67 [11514.08 to 34508.20] | 35536.25 [29386.75 to 59298.64]
  H704_1535_030sN - 50 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_1535_030sN - 50 - 168 |  |  |  |  |  | 20762.95 [15689.00 to 28093.73] | 19437.06 [16763.35 to 22415.96] | 30148.06 [25744.12 to 37295.43] | 18777.41 [13746.93 to 28200.16] | 45959.19 [36503.06 to 107531.61]
  H704_1535_030sN - 80 - 56: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 11 | 12 | 14 | 10 | 13
  H704_1535_030sN - 80 - 56 | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 10.00 [10.00 to 10.00] | 26.97 [26.16 to 28.07] | 10.00 [10.00 to 17.35] | 4856.43 [3691.72 to 5130.60] | 3318.05 [2464.59 to 4052.66] | 6369.54 [5236.11 to 9197.60] | 4460.89 [3900.14 to 6849.22] | 10429.26 [9712.20 to 14126.49]
  H704_1535_030sN - 80 - 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 10 | 9 | 10 | 6
  H704_1535_030sN - 80 - 168 |  |  |  |  |  | 4578.94 [3360.51 to 9386.05] | 3858.60 [3498.92 to 4658.16] | 7070.55 [6571.35 to 8506.66] | 3735.43 [2624.14 to 6140.06] | 14169.87 [12229.59 to 19884.28]

18. Secondary Outcome: Occurrence of Anti-drug Antibodies (ADA) for Participants in Parts A and B
Description: Anti-drug Antibodies (ADA) occurrence in each group measured at prespecified timepoints for all participants in all groups regardless of how many product administrations and how much product they received. Tier 2 responses are only generated for participants who had positive responses to Tier 1.
Time Frame: Measured during Screening, Days 0, 112*, 168†, and 280* Days with † are only available for T1-T5 Days with * are only available for T6-T10
Population: Overall Number of Participants Analyzed represents the number of enrolled participants. Number Analyzed-shows the number of participants with available data after filtering for assay specific quality control criteria at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 16 | 16 | 16 | 16 | 16
Participants
  PGDM1400LS - Tier 1 - 0: number analyzed (Participants) | 3 | 3 | 2 | 3 | 3 | 16 | 16 | 16 | 16 | 16
  PGDM1400LS - Tier 1 - 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0
  PGDM1400LS - Tier 1 - 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  PGDM1400LS - Tier 1 - 112 |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
  PGDM1400LS - Tier 1 - 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
  PGDM1400LS - Tier 1 - 168 | 0 | 0 | 0 | 0 | 0 |  |  |  |  |
  PGDM1400LS - Tier 1 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 15 | 15 | 16 | 14
  PGDM1400LS - Tier 1 - 280 |  |  |  |  |  | 0 | 1 | 0 | 0 | 0
  PGDM1400LS - Tier 2 - 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0
  PGDM1400LS - Tier 2 - 0 |  |  |  |  |  | 1 | 1 | 1 | 2 |
  PGDM1400LS - Tier 2 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PGDM1400LS - Tier 2 - 280 |  |  |  |  |  |  | 1 |  |  |
  PGT121.414.LS - Tier 1 - 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 16 | 16 | 16 | 16 | 16
  PGT121.414.LS - Tier 1 - 0 |  |  |  |  |  | 5 | 6 | 3 | 1 | 3
  PGT121.414.LS - Tier 1 - 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  PGT121.414.LS - Tier 1 - 112 |  |  |  |  |  | 0 | 0 | 0 | 0 | 0
  PGT121.414.LS - Tier 1 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 15 | 15 | 16 | 14
  PGT121.414.LS - Tier 1 - 280 |  |  |  |  |  | 0 | 1 | 0 | 0 | 0
  PGT121.414.LS - Tier 2 - 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 3 | 1 | 3
  PGT121.414.LS - Tier 2 - 0 |  |  |  |  |  | 1 | 3 | 1 | 1 | 1
  PGT121.414.LS - Tier 2 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PGT121.414.LS - Tier 2 - 280 |  |  |  |  |  |  | 0 |  |  |
  VRC07-523LS - Tier 1 - 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 16 | 16 | 16 | 16 | 16
  VRC07-523LS - Tier 1 - 0 |  |  |  |  |  | 1 | 3 | 3 | 4 | 2
  VRC07-523LS - Tier 1 - 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 16 | 16 | 14
  VRC07-523LS - Tier 1 - 112 |  |  |  |  |  | 0 | 1 | 0 | 0 | 0
  VRC07-523LS - Tier 1 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 15 | 15 | 16 | 14
  VRC07-523LS - Tier 1 - 280 |  |  |  |  |  | 0 | 0 | 1 | 2 | 0
  VRC07-523LS - Tier 2 - 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 4 | 2
  VRC07-523LS - Tier 2 - 0 |  |  |  |  |  | 0 | 2 | 1 | 1 | 1
  VRC07-523LS - Tier 2 - 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  VRC07-523LS - Tier 2 - 112 |  |  |  |  |  |  | 0 |  |  |
  VRC07-523LS - Tier 2 - 280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
  VRC07-523LS - Tier 2 - 280 |  |  |  |  |  |  |  | 0 | 0 |

19. Secondary Outcome: Anti-drug Antibodies (ADA) Titers for Participants in Parts A and B
Description: Anti-drug Antibodies (ADA) tier 3 titers in each group measured at prespecified timepoints for all participants in all groups regardless of how many product administrations and how much product they received. Tier 3 titers are only available for those participants who had positive for ADA Tiers 1 and 2.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: titer
Arm/Group | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
Number analyzed (Participants) | 2 | 5 | 2 | 4 | 2
titer
  PGDM1400LS - Tier 3 - 0: number analyzed (Participants) | 1 | 1 | 1 | 2 | 0
  PGDM1400LS - Tier 3 - 0 | 1 [1 to 1] | 243 [243 to 243] | 27 [27 to 27] | 3 [3 to 3] |
  PGDM1400LS - Tier 3 - 280: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  PGDM1400LS - Tier 3 - 280 |  | 3 [3 to 3] |  |  |
  PGT121.414.LS - Tier 3 - 0: number analyzed (Participants) | 1 | 3 | 1 | 1 | 1
  PGT121.414.LS - Tier 3 - 0 | 9 [9 to 9] | 3 [2 to 15] | 2187 [2187 to 2187] | 1 [1 to 1] | 1 [1 to 1]
  VRC07-523LS - Tier 3 - 0: number analyzed (Participants) | 0 | 2 | 1 | 1 | 1
  VRC07-523LS - Tier 3 - 0 |  | 15 [9 to 21] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]

ADVERSE EVENTS:
Time Frame: The study Unsolicited AE reporting time frame is from study enrollment of a trial participant to (and including) Day 168 for T1-T5 and Day 280 for T6-T10. The Solicited AE assessment were collected through 3 full days after each vaccination (vaccinations were given at Day 0 for T1-T5 and Days 0 and 112 for T6-T10)
Arm/Group | T1: PGDM1400LS (IV) 5 mg/kg mo 0 | T2: PGDM1400LS (IV) 20 mg/kg mo 0 | T3: PGDM1400LS (SC) 20 mg/kg mo 0 | T4: PGDM1400LS (IV) 40 mg/kg mo 0 | T5: PGDM1400LS (SC) 40 mg/kg mo 0 | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/3 | 1/3 | 3/3 | 13/16 | 15/16 | 13/16 | 15/16 | 12/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T1: PGDM1400LS (IV) 5 mg/kg mo 0 (N=3) | T2: PGDM1400LS (IV) 20 mg/kg mo 0 (N=3) | T3: PGDM1400LS (SC) 20 mg/kg mo 0 (N=3) | T4: PGDM1400LS (IV) 40 mg/kg mo 0 (N=3) | T5: PGDM1400LS (SC) 40 mg/kg mo 0 (N=3) | T6: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 2 (N=16) | T7: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 2 (N=16) | T8: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) 1 (N=16) | T9: PGDM1400LS + VRC07-523LS + PGT121.414LS (SC) 1 (N=16) | T10: PGDM1400LS + VRC07-523LS + PGT121.414LS (IV) (N=16)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea(Solicited) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Administration site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Administration site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills(Solicited) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (11) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema(Solicited) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 6 (6) | 0 (0)
Infusion site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Infusion site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 2 (3) | 0 (0)
Infusion site pain(Solicited) (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 7 (7) | 3 (3) | 13 (13) | 2 (2)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 2 (4) | 0 (0)
Infusion site swelling(Solicited) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 6 (6) | 0 (0)
Infusion site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise(Solicited) (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 6 (6) | 7 (7) | 5 (5) | 3 (3)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Body temperature increased(Solicited) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia(Solicited) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia(Solicited) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 4 (4) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Headache(Solicited) (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 9 (9) | 6 (6) | 6 (6) | 4 (4) | 6 (6)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea(Solicited) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperhidrosis(Solicited) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pruritus(Solicited) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing(Solicited) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT05184452/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT05184452/SAP_001.pdf